CLINICAL TRIAL: NCT03674112
Title: A Randomized, Multicenter, Open-Label Cross-Over Study to Evaluate Patient Preference and Satisfaction of Subcutaneous Administration of the Fixed-Dose Combination of Pertuzumab and Trastuzumab in Patients With HER2-Positive Early Breast Cancer
Brief Title: A Study to Evaluate Patient Preference and Satisfaction of Subcutaneous Administration of the Fixed-Dose Combination of Pertuzumab and Trastuzumab in Participants With HER2-Positive Early Breast Cancer
Acronym: PHranceSCa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MO40628; 2018-002153-30 (EudraCT Number)
Expanded Access: NCT04395508 (Approved for marketing)
Record Dates: First submitted 2018-09-12; First posted 2018-09-17 (Actual); Results first posted 2021-04-26 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: HER2-Positive Early Breast Cancer
MeSH Terms: interventions — pertuzumab; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- A: P+H IV Followed by PH FDC SC (Experimental): In the Treatment Cross-Over Period of the study, participants randomized to Arm A first received pertuzumab IV and trastuzumab IV (P+H IV) administration for 3 treatment cycles followed by the pertuzumab and trastuzumab fixed-dose combination for subcutaneous administration (PH FDC SC) for 3 treatment cycles (1 cycle = 21 days). Following completion of this study period, participants chose one of the two study treatments to receive in the Treatment Continuation Period for the remaining anti-HER2 treatment cycles (18 planned cycles in total, including pre-study neoadjuvant treatment). After completing study treatment, participants entered the Follow-up Period wherein they were to be followed for 3 years from the date the last participant was randomized.
  Interventions: Drug: Pertuzumab and Trastuzumab Fixed-Dose Combination for Subcutaneous Administration (PH FDC SC); Drug: Pertuzumab IV; Drug: Trastuzumab IV
- B: PH FDC SC Followed by P+H IV (Experimental): In the Treatment Cross-Over Period of the study, participants randomized to Arm B first received the pertuzumab and trastuzumab fixed-dose combination for subcutaneous administration (PH FDC SC) for 3 treatment cycles followed by pertuzumab intravenous (IV) and trastuzumab IV (P+H IV) administration for 3 treatment cycles (1 cycle = 21 days). Following completion of this study period, participants chose one of the two study treatments to receive in the Treatment Continuation Period for the remaining anti-HER2 treatment cycles (18 planned cycles in total, including pre-study neoadjuvant treatment). After completing study treatment, participants entered the Follow-up Period wherein they were to be followed for 3 years from the date the last participant was randomized.
  Interventions: Drug: Pertuzumab and Trastuzumab Fixed-Dose Combination for Subcutaneous Administration (PH FDC SC); Drug: Pertuzumab IV; Drug: Trastuzumab IV

INTERVENTIONS:
Drug: Pertuzumab and Trastuzumab Fixed-Dose Combination for Subcutaneous Administration (PH FDC SC) — PH FDC SC will be administered subcutaneously (SC) at a fixed non-weight-based dose. A loading dose of 1200 mg pertuzumab and 600 mg trastuzumab is then followed by a maintenance dose of 600 mg pertuzumab and 600 mg trastuzumab once every 3 weeks (Q3W).
  Other Names: PH FDC SC; Pertuzumab, Trastuzumab, and Hyaluronidase-zzxf; PHESGO™; RO7198574; RG6264
Drug: Pertuzumab IV — Pertuzumab will be administered intravenously (IV) as a fixed non-weight-based dose of 840-mg IV loading dose and then 420-mg IV maintenance dose Q3W.
  Other Names: Perjeta®
Drug: Trastuzumab IV — Trastuzumab will be administered intravenously (IV) as an 8-mg/kg IV loading dose and then 6 mg/kg IV maintenance dose Q3W.
  Other Names: Herceptin®

SUMMARY:
This is a Phase II, randomized, multicentre, multinational, open-label, cross-over study in adult patients who have completed neoadjuvant chemotherapy with neoadjuvant pertuzumab and trastuzumab and have undergone surgical treatment of human epidermal growth factor receptor 2 (HER2)-positive early breast cancer. The study will consist of two adjuvant treatment periods: a treatment cross-over period and a treatment continuation period. It will evaluate participant-reported preference for a subcutaneously administered fixed-dose combination formulation (FDC SC) of pertuzumab and trastuzumab compared with intravenously (IV) administered pertuzumab and trastuzumab formulations. The study will also evaluate participant-reported satisfaction with pertuzumab and trastuzumab FDC SC and health-related quality of life outcomes; healthcare professionals' perceptions of time/resource use and convenience of pertuzumab and trastuzumab FDC SC compared with pertuzumab and trastuzumab IV formulations; as well as the safety and efficacy of each study regimen.

ELIGIBILITY:
Inclusion Criteria:

Disease-specific criteria:

* Female or male with histologically confirmed, HER2-positive (HER2+) inflammatory, locally advanced or early-stage breast cancer who have received neoadjuvant pertuzumab and trastuzumab and have completed neoadjuvant chemotherapy and subsequently undergone surgery for their breast cancer.
* HER2+ breast cancer assessed at the local laboratory prior to initiation of neoadjuvant therapy. HER2+ status must be determined based on breast biopsy material obtained prior to neoadjuvant treatment and is defined as 3+ by immunohistochemistry (IHC) and/or positive by HER2 amplification by in situ hybridization (ISH) with a ratio of ≥2 for the number of HER2 gene copies to the number of chromosome 17 copies.
* Hormone receptor status of the primary tumour determined by local assessment. Hormone receptor status may be either positive or negative.
* Completed all neoadjuvant chemotherapy and surgery. Adjuvant radiotherapy may be planned or ongoing at study entry and adjuvant hormone therapy is allowed during the study. Note that study treatment cannot be initiated within <2 weeks of surgery but must be initiated ≤9 weeks from the last administration of systemic neoadjuvant therapy.
* No evidence of residual, locally recurrent or metastatic disease after completion of surgery. Patients with clinical suspicion of metastases must undergo radiological assessments per institutional practice to rule out distant disease.
* Wound healing after breast cancer surgery adequate per investigator's assessment to allow initiation of study treatment within ≤9 weeks of last systemic neoadjuvant therapy
* No adjuvant chemotherapy planned. Note that adjuvant hormonal treatment is allowed during the study.

General criteria:

* Ability to comply with the study protocol, in the investigator's judgment
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Intact skin at planned site of subcutaneous injections (thigh)
* Left ventricular ejection fraction (LVEF) ≥55% measured by echocardiogram (ECHO) or multiple-gated acquisition (MUGA) scan within 28 days of study randomization
* No major surgical procedure unrelated to breast cancer within 28 days prior to randomization or anticipation of the need for major surgery during the course of study treatment
* For women of childbearing potential: agreement to remain abstinent or use contraceptive measures, and agreement to refrain from donating eggs, Women must remain abstinent or use non-hormonal contraceptive methods with a failure rate of <1% per year, or two effective non-hormonal contraceptive methods during the study treatment periods and for 7 months after the last dose of study treatment
* For men: agreement to remain abstinent or use a condom, and agreement to refrain from donating sperm, men must remain abstinent or use a condom during the study treatment periods and for seven months after the last dose of study treatment to avoid exposing the embryo. Men must refrain from donating sperm during this same period
* A negative serum pregnancy test must be available prior to randomization for women of childbearing potential

Exclusion Criteria:

Cancer-specific criteria:

* Stage IV (metastatic) breast cancer
* Current or prior history of active malignancy within the last five years. Appropriately treated non-melanoma skin cancer; in situ carcinomas, including cervix, colon, or skin; or Stage I uterine cancer within the last five years are allowed
* Previous systemic therapy for treatment or prevention of breast cancer, except neoadjuvant Perjeta, Herceptin and chemotherapy for current breast cancer

General criteria:

* Investigational treatment within four weeks of enrolment
* Serious cardiac illness or medical conditions
* History of ventricular dysrhythmias or risk factors for ventricular dysrhythmias, such as structural heart disease, coronary heart disease, clinically significant electrolyte abnormalities, or family history of sudden unexplained death or long QT syndrome
* Inadequate bone marrow, renal and impaired liver function
* Current severe, uncontrolled systemic disease that may interfere with planned treatment
* Pregnant or breastfeeding, or intending to become pregnant during the study or within seven months after the last dose of study treatment. Women of childbearing potential must have a negative serum pregnancy test result within seven days prior to initiation of study treatment
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in, and completion of, the study
* Known active liver disease, for example, active viral hepatitis infection, autoimmune hepatic disorders, or sclerosing cholangitis
* Concurrent, serious, uncontrolled infections, or known infection with human immunodeficiency virus (HIV)
* Known hypersensitivity to any of the study drugs, excipients, and/or murine proteins
* Current chronic daily treatment with corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2022-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (40):
- United States (9):
  - Rocky Mountain Cancer Center - Lakewood (West), Lakewood, Colorado
  - Illinois Cancer Care, Peoria, Illinois
  - Cancer Center of Kansas, Wichita, Kansas
  - Maryland Oncology Hematology, Rockville, Maryland
  - Texas Oncology - Dallas Presbyterian Hospital, Dallas, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - Memorial City, Houston, Texas
  - USOR - Texas Oncology - San Antonio Northeast, San Antonio, Texas
  - Texas Oncology- Northeast Texas, Tyler, Texas
- Hospital Britanico de Buenos Aires, Ciudad Autonoma Buenos Aires, Argentina
- Brazil (4):
  - Instituto de Câncer E Transplante, Curitiba, Paraná
  - Clinicas Oncologicas Integradas - COI, Rio de Janeiro, Rio de Janeiro
  - Instituto de Ensino e Pesquisa Sao Lucas - IEP, São Paulo, São Paulo
  - Núcleo de Pesquisa São Camilo; ONCOLOGIA CLINICA / QUIMIOTERAPIA, São Paulo, São Paulo
- Bradford Hill Centro de Investigaciones Clinicas, Recoleta, Chile
- Cuba (2):
  - Hospital Hermanos Ameijeiras, La Habana
  - Instituto Nacional de Oncología y Radiología (INOR), La Habana
- Finland (2):
  - KYS Sadesairaala; Syopatautien poliklinikka, Kuopio
  - VAASAN KESKUSSAIRAALA; Onkologian poliklinikka, Vaasa
- Hong Kong (2):
  - Princess Margaret Hospital, Oncology; Department of Oncology, Hong Kong
  - Prince of Wales Hosp; Dept. Of Clinical Onc, Shatin
- King Hussein Cancer Center, Amman, Jordan
- Lebanon (2):
  - Bellevue Medical Center, El-Metn
  - Hammoud Hospital, Saida
- Mexico (3):
  - Consultorio Privado (José Luis González Trujillo), León, Guanajuato
  - Centro Médico Zambrano Hellion, Monterrey, Nuevo León
  - Cuidados oncologicos, Querétaro City, Querétaro
- Panama (2):
  - Centro Oncológico de Panamá, Panama City
  - Centro Hemato Oncologico Panama, Panama City
- Portugal (3):
  - Hospital da Luz; Departamento de Oncologia Medica, Lisbon
  - Hospital de Santa Maria; Servico de Oncologia Medica, Lisbon
  - IPO do Porto; Servico de Oncologia Medica, Porto
- National Center for Cancer Care and Research, Doha, Qatar
- King Fahad Medical City; Gastroentrology, Riyadh, Saudi Arabia
- Serbia (2):
  - Institute of Oncology and Radiology of Serbia, Belgrade
  - Clinical Centre Nis, Clinic for Oncology, Niš
- Spain (2):
  - Hospital General Universitario de Elche; Servicio de Oncologia, Elche, Alicante
  - Hospital Universitario de Canarias;servicio de Oncologia, San Cristóbal de La Laguna, Tenerife
- Sweden (2):
  - Sodersjukhuset; Onkologkliniken, Stockholm
  - Västmanlands sjukhus Västerås, Onkologkliniken, Västerås

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/).
  For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] O'Shaughnessy J, Sousa S, Cruz J, Fallowfield DL, Auvinen P, Pulido C, Cvetanovic A, Wilks S, Ribeiro L, Burotto M, Boulet T, Revelant V, Theron N, Trask P, Wahyudi L, Kirchmayer Machackova Z, Stamatovic L. Long-Term Safety and Efficacy of the Fixed-Dose Combination of Pertuzumab and Trastuzumab for Subcutaneous Injection in Patients With HER2-Positive Early Breast Cancer in PHranceSCa, a Randomized, Open-Label Phase II Study. Clin Breast Cancer. 2025 Aug;25(6):554-559.e1. doi: 10.1016/j.clbc.2025.04.016. Epub 2025 May 3. PMID 40461387
- [Derived] O'Shaughnessy J, Sousa S, Cruz J, Fallowfield L, Auvinen P, Pulido C, Cvetanovic A, Wilks S, Ribeiro L, Burotto M, Klingbiel D, Messeri D, Alexandrou A, Trask P, Fredriksson J, Machackova Z, Stamatovic L; PHranceSCa study group. Preference for the fixed-dose combination of pertuzumab and trastuzumab for subcutaneous injection in patients with HER2-positive early breast cancer (PHranceSCa): A randomised, open-label phase II study. Eur J Cancer. 2021 Jul;152:223-232. doi: 10.1016/j.ejca.2021.03.047. Epub 2021 Jun 16. PMID 34147014

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 183 patients were screened and 160 participants were enrolled.
Period: Treatment Cross-Over (Cycles 1 to 6)
Arm/Group | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Started | 80 | 80
Completed Cross-Over Treatment (Received all 6 cycles of cross-over treatment) | 80 | 80
Completed (Completed the Treatment Cross-Over Period) | 79 (One participant discontinued the cross-over period after completing cross-over treatment (after receiving Cycle 6) and did not start treatment continuation. They entered directly into the follow-up period.) | 80
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Treatment Continuation (Cycles 7 to ≤18)
Arm/Group | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Started | 79 | 80
Received PH FDC SC for Treatment Continuation | 70 | 68
Received P+H IV for Treatment Continuation | 9 | 12
Completed Continuation Treatment (Received all cycles of continuation treatment (from Cycle 7 up to 18 total cycles of neo/adjuvant treatment)) | 78 | 77 (One participant withdrew from the study during the continuation period (withdrawal by subject) and did not enter follow-up.)
Completed (Completed the Treatment Continuation Period) | 78 | 77
Not Completed | 1 | 3
Not completed — Reason Not Specified | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Disease Relapse | 1 | 0
Period: Follow-Up Period (≥3 Years)
Arm/Group | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Started (Participants who discontinued previous treatment periods but remained in the study continued into the follow-up period.) | 80 | 79
Completed | 73 | 75
Not Completed | 7 | 4
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Death | 2 | 0
Not completed — Reason Not Specified | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: includes all randomized participants, allocated to their randomized treatment arm, whether or not the assigned study treatment was received.
Groups:
- Total: Total of all reporting groups
Arm/Group | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.4 (11.6) | 48.2 (12.1) | 48.8 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 80 | 160
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 21 | 38
  Not Hispanic or Latino | 59 | 54 | 113
  Unknown or Not Reported | 4 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 3 | 8
  Asian | 8 | 4 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 62 | 67 | 129
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 7
Baseline Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 67.36 (12.08) | 70.21 (14.15) | 68.78 (13.20)
Eastern Cooperative Oncology Group (ECOG) Performance Status at Baseline [Count of Participants; unit: Participants] — ECOG Performance Status: 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework or office work.
  Participants
    ECOG Peformance Status 0 | 70 | 70 | 140
    ECOG Peformance Status 1 | 10 | 10 | 20
Number of Cycles of Prior Neoadjuvant Pertuzumab IV and Trastuzumab IV [Count of Participants; unit: Participants]
  <4 Cycles | 5 | 10 | 15
  ≥4 Cycles | 75 | 70 | 145
Prior Neoadjuvant Chemotherapy Regimen [Count of Participants; unit: Participants] — Participants were stratified at randomization according to prior neoadjuvant chemotherapy regimen, pathological complete response to prior neoadjuvant treatment, and hormone receptor status.
  Participants
    Anthracyclines + Taxanes | 55 | 53 | 108
    Carboplatin + Taxanes | 22 | 23 | 45
    Taxanes Only | 3 | 4 | 7
Pathological Complete Response (pCR) to Prior Neoadjuvant Treatment [Count of Participants; unit: Participants] — Participants were stratified at randomization according to prior neoadjuvant chemotherapy regimen, pathological complete response to prior neoadjuvant treatment, and hormone receptor status.
  Participants
    pCR | 52 | 50 | 102
    Non-pCR | 28 | 30 | 58
Hormone Receptor Status [Count of Participants; unit: Participants] — Participants were stratified at randomization according to prior neoadjuvant chemotherapy regimen, pathological complete response to prior neoadjuvant treatment, and hormone receptor status.
  Participants
    Estrogen Receptor (ER)-Positive and/or Progesterone Receptor (PgR)-Positive | 53 | 51 | 104
    ER-Negative and PgR-Negative | 27 | 29 | 56

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants by Their Preferred Method of Pertuzumab and Trastuzumab Administration, as Assessed in Question 1 of the Patient Preference Questionnaire (PPQ)
Description: Question 1 of the Patient Preference Questionnaire (PPQ) asked participants the following question: "All things considered, which method of administration did you prefer?" The three available options for a participant's response were: IV, SC, or No preference. A point estimate with associated exact Clopper-Pearson binomial 95% confidence interval was calculated only for the percentage of participants who preferred PH FDC SC.
Time Frame: Cycle 6 Day 1 (each cycle is 21 days)
Population: Modified Intent-to-Treat (mITT) Population: All randomized participants, allocated to their randomized treatment arm, who received at least one dose by both SC and IV routes of administration during the Treatment Cross-over Period and subsequently answered at least Question 1 of the PPQ.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- All Participants: In the Treatment Cross-Over Period of the study, all participants received their first 6 cycles of treatment in accordance with the study arm to which they were randomized: Arm A) pertuzumab IV and trastuzumab IV (P+H IV) for 3 treatment cycles followed by the pertuzumab and trastuzumab fixed-dose combination for subcutaneous administration (PH FDC SC) for 3 treatment cycles (1 cycle = 21 days); or Arm B) PH FDC SC for 3 treatment cycles followed by P+H IV for 3 treatment cycles (1 cycle = 21 days). Following completion of this study period, participants chose one of the two study treatments to receive in the Treatment Continuation Period for the remaining anti-HER2 treatment cycles (18 planned cycles in total, including pre-study neoadjuvant treatment). After completing study treatment, participants entered the Follow-up Period wherein they were to be followed for 3 years from the date the last participant was randomized.
Arm/Group | All Participants | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 160 | 80 | 80
Percentage of participants
  SC Preference | 85.00 [78.51 to 90.15] | 87.50 [78.21 to 93.84] | 82.50 [72.38 to 90.09]
  IV Preference | 13.8 [NA to NA] — As per the statistical analysis plan, a 95% confidence interval was only calculated for the percentage of participants who preferred PH FDC SC. | 12.5 [NA to NA] — As per the statistical analysis plan, a 95% confidence interval was only calculated for the percentage of participants who preferred PH FDC SC. | 15.0 [NA to NA] — As per the statistical analysis plan, a 95% confidence interval was only calculated for the percentage of participants who preferred PH FDC SC.
  No Preference | 1.3 [NA to NA] — As per the statistical analysis plan, a 95% confidence interval was only calculated for the percentage of participants who preferred PH FDC SC. | 0.0 [NA to NA] — As per the statistical analysis plan, a 95% confidence interval was only calculated for the percentage of participants who preferred PH FDC SC. | 2.5 [NA to NA] — As per the statistical analysis plan, a 95% confidence interval was only calculated for the percentage of participants who preferred PH FDC SC.

2. Secondary Outcome: Percentage of Participants by Responses to the Strength of Their Preferred Method of Pertuzumab and Trastuzumab Administration, as Assessed in Question 2 of the Patient Preference Questionnaire (PPQ)
Description: Question 1 of the Patient Preference Questionnaire (PPQ) was as follows: "All things considered, which method of administration did you prefer?" The available options for a participant's response were IV, SC, or No preference. In Question 2 of the PPQ, participants who reported a preference for one of the two administration routes in Question 1 of the PPQ were asked to rate the strength of their preference (very strong, fairly strong, not very strong).
Time Frame: Cycle 6 Day 1 (each cycle is 21 days)
Population: Modified ITT (mITT) Population; for Question 2 of the PPQ, the number analyzed for the strength of SC or IV preference represents the participants who indicated in their responses to Question 1 of the PPQ that they preferred the SC or IV route of administration, respectively.
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 158 | 80 | 78
Percentage of participants
  SC Preference: Very Strong: number analyzed (Participants) | 136 | 70 | 66
  SC Preference: Very Strong | 67.6 | 68.6 | 66.7
  SC Preference: Fairly Strong: number analyzed (Participants) | 136 | 70 | 66
  SC Preference: Fairly Strong | 25.0 | 24.3 | 25.8
  SC Preference: Not Very Strong: number analyzed (Participants) | 136 | 70 | 66
  SC Preference: Not Very Strong | 7.4 | 7.1 | 7.6
  IV Preference: Very Strong: number analyzed (Participants) | 22 | 10 | 12
  IV Preference: Very Strong | 54.5 | 40.0 | 66.7
  IV Preference: Fairly Strong: number analyzed (Participants) | 22 | 10 | 12
  IV Preference: Fairly Strong | 9.1 | 10.0 | 8.3
  IV Preference: Not Very Strong: number analyzed (Participants) | 22 | 10 | 12
  IV Preference: Not Very Strong | 36.4 | 50.0 | 25.0

3. Secondary Outcome: Percentage of Responses From Participants to the Two Main Reasons for Their Preferred Method of Pertuzumab and Trastuzumab Administration, as Assessed in Question 3 of the Patient Preference Questionnaire (PPQ)
Description: In Question 3 of the PPQ, participants who reported a preference for one of the two administration routes in Question 1 of the PPQ were asked to provide the two main reasons for their preference. The five available options for a participant's response were: Feels less emotionally distressing; Requires less time in the clinic; Lower level of injection-site pain; Feels more comfortable during administration; and Other reason.
Time Frame: Cycle 6 Day 1 (each cycle is 21 days)
Population: Modified ITT (mITT) Population; for Question 3, the number analyzed for the two main reasons for SC or IV preference represents the participants who indicated in their responses to Question 1 of the PPQ that they preferred the SC or IV route of administration, respectively.
Measure: Number; unit: Percentage of responses
Units Other Than Participants: Responses
Arm/Group | All Participants | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 158 | 80 | 78
Number analyzed (Responses) | 324 | 160 | 164
Percentage of responses
  SC Preference: Feels Less Emotionally Distressing: number analyzed (Participants) | 136 | 70 | 66
  SC Preference: Feels Less Emotionally Distressing: number analyzed (Responses) | 282 | 143 | 139
  SC Preference: Feels Less Emotionally Distressing | 16.3 | 14.7 | 18.0
  SC Preference: Requires Less Time in the Clinic: number analyzed (Participants) | 136 | 70 | 66
  SC Preference: Requires Less Time in the Clinic: number analyzed (Responses) | 282 | 143 | 139
  SC Preference: Requires Less Time in the Clinic | 42.2 | 42.0 | 42.4
  SC Preference: Lower Level of Injection-Site Pain: number analyzed (Participants) | 136 | 70 | 66
  SC Preference: Lower Level of Injection-Site Pain: number analyzed (Responses) | 282 | 143 | 139
  SC Preference: Lower Level of Injection-Site Pain | 11.3 | 9.8 | 12.9
  SC Preference: Feels More Comfortable During Administration: number analyzed (Participants) | 136 | 70 | 66
  SC Preference: Feels More Comfortable During Administration: number analyzed (Responses) | 282 | 143 | 139
  SC Preference: Feels More Comfortable During Administration | 25.9 | 28.7 | 23.0
  SC Preference: Other Reason: number analyzed (Participants) | 136 | 70 | 66
  SC Preference: Other Reason: number analyzed (Responses) | 282 | 143 | 139
  SC Preference: Other Reason | 4.3 | 4.9 | 3.6
  IV Preference: Feels Less Emotionally Distressing: number analyzed (Participants) | 22 | 10 | 12
  IV Preference: Feels Less Emotionally Distressing: number analyzed (Responses) | 42 | 17 | 25
  IV Preference: Feels Less Emotionally Distressing | 16.7 | 17.6 | 16.0
  IV Preference: Requires Less Time in the Clinic: number analyzed (Participants) | 22 | 10 | 12
  IV Preference: Requires Less Time in the Clinic: number analyzed (Responses) | 42 | 17 | 25
  IV Preference: Requires Less Time in the Clinic | 4.8 | 5.9 | 4.0
  IV Preference: Lower Level of Injection-Site Pain: number analyzed (Participants) | 22 | 10 | 12
  IV Preference: Lower Level of Injection-Site Pain: number analyzed (Responses) | 42 | 17 | 25
  IV Preference: Lower Level of Injection-Site Pain | 26.2 | 23.5 | 28.0
  IV Preference: Feels More Comfortable During Administration: number analyzed (Participants) | 22 | 10 | 12
  IV Preference: Feels More Comfortable During Administration: number analyzed (Responses) | 42 | 17 | 25
  IV Preference: Feels More Comfortable During Administration | 33.3 | 47.1 | 24.0
  IV Preference: Other Reason: number analyzed (Participants) | 22 | 10 | 12
  IV Preference: Other Reason: number analyzed (Responses) | 42 | 17 | 25
  IV Preference: Other Reason | 19.0 | 5.9 | 28.0

4. Secondary Outcome: Percentage of Participants by Their Level of Satisfaction With the Respective Methods of Administration (IV and SC), Question 1 of the Therapy Administration Satisfaction Questionnaire -Intravenous (TASQ-IV) and -Subcutaneous (TASQ-SC)
Description: The Therapy Administration Satisfaction Questionnaire (TASQ) is a 12-item, patient-reported questionnaire measuring the impact of each mode of treatment administration (TASQ-IV for IV treatment and TASQ-SC for SC treatment) on five domains: Physical Impact, Psychological Impact, Impact on Activities of Daily Living, Convenience, and Satisfaction. The TASQ-IV/-SC was administered at treatment Cycles 3 and 6 according to the order of treatment received per arm during the Cross-Over Period. Question 1 of the TASQ-IV/TASQ-SC is one of two items in the Satisfaction domain, with participants providing their answers to the following question: "How satisfied or dissatisfied were you with the IV infusion/SC injection?" The five available options for a participant's response were: very satisfied, satisfied, neither satisfied nor dissatisfied, dissatisfied, and very dissatisfied.
Time Frame: Cycle 3 Day 1, Cycle 6 Day 1 (each cycle is 21 days)
Population: Modified Intent-to-Treat (mITT) Population
Measure: Number; unit: Percentage of participants
Groups:
- All Participants: TASQ-IV Completers: This analysis set includes all participants from Arms A and B who completed the TASQ-IV questionnaire, which was administered at the last IV treatment cycle in the Treatment Cross-Over Period of the study. During the Treatment Cross-Over Period, all participants received their first 6 cycles of treatment in accordance with the study arm to which they were randomized: Arm A) pertuzumab IV and trastuzumab IV (P+H IV) for 3 treatment cycles followed by the pertuzumab and trastuzumab fixed-dose combination for subcutaneous administration (PH FDC SC) for 3 treatment cycles (1 cycle = 21 days); or Arm B) PH FDC SC for 3 treatment cycles followed by P+H IV for 3 treatment cycles (1 cycle = 21 days). Following completion of this study period, participants chose one of the two study treatments to receive in the Treatment Continuation Period for the remaining anti-HER2 treatment cycles (18 planned cycles in total, including pre-study neoadjuvant treatment). After completing study treatment, participants entered the Follow-up Period wherein they were to be followed for 3 years from the date the last participant was randomized.
- All Participants: TASQ-SC Completers: This analysis set includes all participants from Arms A and B who completed the TASQ-SC questionnaire, which was administered at the last SC treatment cycle in the Treatment Cross-Over Period of the study. During the Treatment Cross-Over Period, all participants received their first 6 cycles of treatment in accordance with the study arm to which they were randomized: Arm A) pertuzumab IV and trastuzumab IV (P+H IV) for 3 treatment cycles followed by the pertuzumab and trastuzumab fixed-dose combination for subcutaneous administration (PH FDC SC) for 3 treatment cycles (1 cycle = 21 days); or Arm B) PH FDC SC for 3 treatment cycles followed by P+H IV for 3 treatment cycles (1 cycle = 21 days). Following completion of this study period, participants chose one of the two study treatments to receive in the Treatment Continuation Period for the remaining anti-HER2 treatment cycles (18 planned cycles in total, including pre-study neoadjuvant treatment). After completing study treatment, participants entered the Follow-up Period wherein they were to be followed for 3 years from the date the last participant was randomized.
Arm/Group | All Participants: TASQ-IV Completers | All Participants: TASQ-SC Completers
Number analyzed (Participants) | 160 | 160
Percentage of participants
  Very Satisfied | 25.6 | 57.5
  Satisfied | 41.9 | 30.6
  Neither Satisfied nor Dissatisfied | 25.6 | 4.4
  Dissatisfied | 5.6 | 1.9
  Very Dissatisfied | 1.3 | 4.4
  Did Not Answer Question | 0.0 | 1.3

5. Secondary Outcome: Mean Scores of the Five Domains of the TASQ-IV and TASQ-SC (Satisfaction, Physical Impact, Psychological Impact, Impact on Activities of Daily Living, and Convenience) to Assess the Impact of IV and SC Routes of Administration
Description: The TASQ is a 12-item, patient-reported questionnaire measuring the impact of the mode of treatment administration (TASQ-IV for IV treatment and TASQ-SC for SC treatment) on 5 domains: Physical Impact (3 items: Question [Q]2. Pain, Q3. Swelling, Q4. Redness), Psychological Impact (1 item: Q5. Feeling restricted), Impact on Activities of Daily Living (1 item: Q8. Lost/gained time), Convenience (2 items: Q6. Is it convenient?, Q7. Bothered by the amount of time?), and Satisfaction (2 items: Q1. How satisfied or dissatisfied are you with treatment?, Q12: Would you recommend the way you received the treatment?). In addition, 3 questions in the TASQ (Q9, Q10, Q11) are not part of the domains. Responses for the 3 domains that contain more than 1 item were scored from 0 to 100, with a higher score indicating a better outcome. Responses for the 2 domains with 1 item were scored from 1 to 5, with a higher score indicating a better outcome.
Time Frame: Cycle 3 Day 1, Cycle 6 Day 1 (each cycle is 21 days)
Population: Modified Intent-to-Treat (mITT) Population; The number analyzed indicates the number of participants who completed the TASQ-IV/-SC questionnaire items within a domain.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | All Participants: TASQ-IV Completers | All Participants: TASQ-SC Completers
Number analyzed (Participants) | 160 | 160
Score on a scale
  Satisfaction Domain: number analyzed (Participants) | 156 | 157
  Satisfaction Domain | 64.3 (23.6) | 87.7 (17.5)
  Physical Impact Domain: number analyzed (Participants) | 159 | 157
  Physical Impact Domain | 86.5 (14.8) | 81.3 (15.4)
  Psychological Impact Domain: number analyzed (Participants) | 160 | 157
  Psychological Impact Domain | 3.8 (1.2) | 4.6 (0.7)
  Impact on Activities of Daily Living Domain: number analyzed (Participants) | 160 | 156
  Impact on Activities of Daily Living Domain | 2.3 (0.9) | 3.9 (1.0)
  Convenience Domain: number analyzed (Participants) | 159 | 157
  Convenience Domain | 56.8 (26.0) | 90.0 (13.8)

6. Secondary Outcome: Percentage of Participants by Their Responses to Question 9 of the TASQ-IV and TASQ-SC, Assessing Whether Participants Receiving IV and SC Administration Have as Much Time as They Would Like to Talk to Their Nurse and/or Doctor About Their Illness
Description: The TASQ is a 12-item, patient-reported questionnaire measuring the impact of the mode of treatment administration (TASQ-IV for IV treatment and TASQ-SC for SC treatment) on 5 domains. In addition, 3 questions (Q.9-11) are not part of the domains. The TASQ-IV/-SC was administered at treatment Cycles 3 and 6 according to the order of treatment received per arm during the Cross-Over Period. Question 9 asked the participant, "When you receive the IV infusion/SC injection treatment, are you able to talk to your nurse and/or doctor as much as you would like about your illness?" There were five available response options: a) Yes, I had more than enough time to talk to my nurse and/or doctor; b) Yes, but I would have liked more time to talk to my nurse and/or doctor; c) It does not matter to me if I have time to talk to my nurse and/or doctor during my treatment; d) No, I did not have enough time to talk to my nurse and/or doctor; and e) No, I did not talk to my nurse and/or doctor at all.
Time Frame: Cycle 3 Day 1 and Cycle 6 Day 1 (each cycle is 21 days)
Population: Modified Intent-to-Treat (mITT) Population
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants: TASQ-IV Completers | All Participants: TASQ-SC Completers
Number analyzed (Participants) | 160 | 160
Percentage of participants
  a) Yes, I had enough time to talk to my nurse and/or doctor | 82.5 | 90.0
  b) Yes, but I would have liked more time to talk to my nurse and/or doctor | 9.4 | 5.0
  c) It does not matter to me if I have time to talk to my nurse and/or doctor | 5.0 | 3.1
  d) No, I did not have enough time to talk to my nurse and/or doctor | 0.6 | 0.6
  e) No, I did not talk to my nurse and/or doctor at all | 2.5 | 0.0
  Patient did not answer question | 0.0 | 1.3

7. Secondary Outcome: Percentage of Participants by Their Responses to Question 10 of the TASQ-IV and TASQ-SC, Assessing Whether IV and SC Administration Have an Impact on the Amount of Time Participants Have to Talk to Their Nurse and/or Doctor About Their Illness
Description: The Therapy Administration Satisfaction Questionnaire (TASQ) is a 12-item, patient-reported questionnaire measuring the impact of the mode of treatment administration (TASQ-IV for IV treatment and TASQ-SC for SC treatment) on 5 domains (questions [Q] 1 to 8 and Q12): Physical Impact, Psychological Impact, Impact on Activities of Daily Living, Convenience, and Satisfaction. In addition, 3 questions in the TASQ-IV/-SC (Q 9-11) are not part of the domains. The TASQ-IV/-SC were administered at treatment Cycles 3 and 6 according to the order of treatment received in each study arm during the Cross-Over Period. Question 10 of the TASQ-IV/-SC asked the participant "Does the IV infusion/SC injection impact the amount of time you have to talk to your nurse and/or doctor about your illness and other concerns?" There were two available options for the participant's response: Yes or No.
Time Frame: Cycle 3 Day 1 and Cycle 6 Day 1 (each cycle is 21 days)
Population: Modified Intent-to-Treat (mITT) Population
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants: TASQ-IV Completers | All Participants: TASQ-SC Completers
Number analyzed (Participants) | 160 | 160
Percentage of participants
  Yes | 20.0 | 13.1
  No | 79.4 | 85.0
  Patient Did Not Answer Question | 0.6 | 1.9

8. Secondary Outcome: Percentage of Participants by Their Responses to Question 11 of the TASQ-IV and TASQ-SC, Assessing the Participants' Preferred Method for Receiving Cancer Treatment
Description: The Therapy Administration Satisfaction Questionnaire (TASQ) is a 12-item, patient-reported questionnaire measuring the impact of the mode of treatment administration (TASQ-IV for IV treatment and TASQ-SC for SC treatment) on 5 domains (questions [Q] 1 to 8 and Q12): Physical Impact, Psychological Impact, Impact on Activities of Daily Living, Convenience, and Satisfaction. In addition, 3 questions in the TASQ-IV/-SC (Q 9-11) are not part of the domains. The TASQ-IV/-SC was administered at treatment Cycles 3 and 6 according to the order of treatment received during the Cross-Over Period. Question 11 of the TASQ-IV/-SC asked the participant, "There are two ways to get cancer treatment: a) IV infusion given through a port or small tube; b) SC (subcutaneous) injection in your thigh. Which would you prefer?" There were three available options for the participant's response: IV, SC, or No Preference.
Time Frame: Cycle 3 Day 1 and Cycle 6 Day 1 (each cycle is 21 days)
Population: Modified Intent-to-Treat (mITT) Population
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants: TASQ-IV Completers | All Participants: TASQ-SC Completers
Number analyzed (Participants) | 160 | 160
Percentage of participants
  Prefer IV Method | 11.9 | 9.4
  Prefer SC Method | 70.6 | 82.5
  No Preference | 11.9 | 5.6
  Patient Did Not Answer Question | 5.6 | 2.5

9. Secondary Outcome: Percentage of Participants by Their Choice of Treatment in the Treatment Continuation Period (PH FDC SC or P+H IV) and by Consistency of This Choice With Their Preferred Method of Administration Reported in Question 1 of the PPQ
Description: At treatment Cycle 6, Day 1, participants were expected to select the study treatment formulation (PH FDC SC or P+H IV) they would receive during the Treatment Continuation Period (starting at Cycle 7) to complete their 18 cycles of neo/adjuvant HER2-targeted treatment. Additionally, for each participant's preference category (SC, IV, and No preference) as per the question 1 of the patient preference questionnaire (PPQ), the percentage of participants who selected each treatment administration route for the Treatment Continuation Period (PH FDC SC or P+H IV) was summarized.
Time Frame: Cycle 6 Day 1 (each cycle is 21 days)
Population: All randomized participants, allocated to their randomized treatment arm.
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 160 | 80 | 80
Percentage of participants
  Chose PH FDC SC for Treatment Continuation | 86.9 | 88.8 | 85.0
  Chose P+H IV for Treatment Continuation | 13.1 | 11.3 | 15.0
  Preferred SC per the PPQ and Chose PH FDC SC for Continuation | 85.0 | 87.5 | 82.5
  Preferred SC per the PPQ and Chose P+H IV for Continuation | 0.0 | 0.0 | 0.0
  Preferred IV per the PPQ and Chose PH FDC SC for Continuation | 0.6 | 1.3 | 0.0
  Preferred IV per the PPQ and Chose P+H IV for Continuation | 13.1 | 11.3 | 15.0
  No Preference per the PPQ and Chose PH FDC SC for Continuation | 1.3 | 0.0 | 2.5
  No Preference per the PPQ and Chose P+H IV for Continuation | 0.0 | 0.0 | 0.0

10. Secondary Outcome: Duration of Treatment Administration Activities According to Healthcare Professionals' Responses on Perception of Time by Treatment Cycle, Question 1 of the Healthcare Professional Questionnaire (HCPQ) - Treatment Room
Description: The Healthcare Professional Questionnaire (HCPQ)-Treatment Room Question 1 was completed at each treatment cycle of the Treatment Cross-Over Period by the healthcare professionals (HCPs) who administered treatment to the study's participants. HCPs responded to the following parts of Question 1 that sought to evaluate the amount of time it took to complete activities related to treatment administration: "If new IV access was needed for this cycle of treatment, please indicate what type of IV access was provided (central venous catheter, peripherally inserted central catheter, or peripheral vein cannulation) and how long (in minutes) this took to set up (only for participants receiving IV treatment)? How long (in minutes) did it take to administer the treatment, i.e. total infusion duration? How long (in minutes) was the patient in the Treatment Room for in total?"
Time Frame: Day 1 of Cycles 1-6 (each cycle is 21 days)
Population: The number analyzed includes HCPs who completed question 1 of the survey per treatment cycle. For the questions related to IV access, the number analyzed only includes HCP responses for participants who required new IV access at a given treatment cycle.
Measure: Median (Full Range); unit: minutes
Arm/Group | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 80 | 80
minutes
  Cycle 1. Duration of Central Venous Catheter Set Up (IV Only)?: number analyzed (Participants) | 4 | 0
  Cycle 1. Duration of Central Venous Catheter Set Up (IV Only)? | 5.0 [4 to 6] |
  Cycle 1. Duration of Peripherally Inserted Central Catheter Set Up (IV Only)?: number analyzed (Participants) | 1 | 0
  Cycle 1. Duration of Peripherally Inserted Central Catheter Set Up (IV Only)? | 5.0 [5 to 5] |
  Cycle 1. Duration of Peripheral Vein Cannulation Set Up (IV Only)?: number analyzed (Participants) | 50 | 0
  Cycle 1. Duration of Peripheral Vein Cannulation Set Up (IV Only)? | 5.0 [1 to 40] |
  Cycle 1. How Long Did it Take to Administer the Treatment?: number analyzed (Participants) | 79 | 79
  Cycle 1. How Long Did it Take to Administer the Treatment? | 150.0 [60 to 396] | 8.0 [2 to 17]
  Cycle 1. How Long Was the Patient in the Treatment Room in Total?: number analyzed (Participants) | 79 | 79
  Cycle 1. How Long Was the Patient in the Treatment Room in Total? | 300.0 [90 to 450] | 50.0 [8 to 240]
  Cycle 2. Duration of Central Venous Catheter Set Up (IV Only)?: number analyzed (Participants) | 4 | 0
  Cycle 2. Duration of Central Venous Catheter Set Up (IV Only)? | 5.0 [3 to 5] |
  Cycle 2. Duration of Peripherally Inserted Central Catheter Set Up (IV Only)?: number analyzed (Participants) | 1 | 0
  Cycle 2. Duration of Peripherally Inserted Central Catheter Set Up (IV Only)? | 3.0 [3 to 3] |
  Cycle 2. Duration of Peripheral Vein Cannulation Set Up (IV Only)?: number analyzed (Participants) | 48 | 0
  Cycle 2. Duration of Peripheral Vein Cannulation Set Up (IV Only)? | 5.0 [1 to 20] |
  Cycle 2. How Long Did it Take to Administer the Treatment?: number analyzed (Participants) | 77 | 80
  Cycle 2. How Long Did it Take to Administer the Treatment? | 90.0 [8 to 260] | 8.0 [5 to 20]
  Cycle 2. How Long Was the Patient in the Treatment Room in Total?: number analyzed (Participants) | 77 | 78
  Cycle 2. How Long Was the Patient in the Treatment Room in Total? | 153.0 [30 to 342] | 40.0 [8 to 225]
  Cycle 3. Duration of Central Venous Catheter Set Up (IV Only)?: number analyzed (Participants) | 5 | 0
  Cycle 3. Duration of Central Venous Catheter Set Up (IV Only)? | 5.0 [3 to 10] |
  Cycle 3. Duration of Peripherally Inserted Central Catheter Set Up (IV Only)?: number analyzed (Participants) | 1 | 0
  Cycle 3. Duration of Peripherally Inserted Central Catheter Set Up (IV Only)? | 3.0 [3 to 3] |
  Cycle 3. Duration of Peripheral Vein Cannulation Set Up (IV Only)?: number analyzed (Participants) | 48 | 0
  Cycle 3. Duration of Peripheral Vein Cannulation Set Up (IV Only)? | 5.0 [1 to 30] |
  Cycle 3. How Long Did it Take to Administer the Treatment?: number analyzed (Participants) | 79 | 80
  Cycle 3. How Long Did it Take to Administer the Treatment? | 70.0 [30 to 240] | 7.5 [4 to 16]
  Cycle 3. How Long Was the Patient in the Treatment Room in Total?: number analyzed (Participants) | 79 | 79
  Cycle 3. How Long Was the Patient in the Treatment Room in Total? | 150.0 [105 to 330] | 36.0 [5 to 327]
  Cycle 4. Duration of Central Venous Catheter Set Up (IV Only)?: number analyzed (Participants) | 0 | 7
  Cycle 4. Duration of Central Venous Catheter Set Up (IV Only)? |  | 5.0 [2 to 10]
  Cycle 4. Duration of Peripherally Inserted Central Catheter Set Up (IV Only)?: number analyzed (Participants) | 0 | 1
  Cycle 4. Duration of Peripherally Inserted Central Catheter Set Up (IV Only)? |  | 42.0 [42 to 42]
  Cycle 4. Duration of Peripheral Vein Cannulation Set Up (IV Only)?: number analyzed (Participants) | 0 | 36
  Cycle 4. Duration of Peripheral Vein Cannulation Set Up (IV Only)? |  | 5.0 [1 to 20]
  Cycle 4. How Long Did it Take to Administer the Treatment?: number analyzed (Participants) | 80 | 77
  Cycle 4. How Long Did it Take to Administer the Treatment? | 8.0 [4 to 12] | 60.0 [30 to 210]
  Cycle 4. How Long Was the Patient in the Treatment Room in Total?: number analyzed (Participants) | 78 | 77
  Cycle 4. How Long Was the Patient in the Treatment Room in Total? | 45.0 [1 to 185] | 150.0 [80 to 480]
  Cycle 5. Duration of Central Venous Catheter Set Up (IV Only)?: number analyzed (Participants) | 0 | 5
  Cycle 5. Duration of Central Venous Catheter Set Up (IV Only)? |  | 3.0 [2 to 10]
  Cycle 5. Duration of Peripherally Inserted Central Catheter Set Up (IV Only)?: number analyzed (Participants) | 0 | 1
  Cycle 5. Duration of Peripherally Inserted Central Catheter Set Up (IV Only)? |  | 10.0 [10 to 10]
  Cycle 5. Duration of Peripheral Vein Cannulation Set Up (IV Only)?: number analyzed (Participants) | 0 | 38
  Cycle 5. Duration of Peripheral Vein Cannulation Set Up (IV Only)? |  | 5.0 [1 to 20]
  Cycle 5. How Long Did it Take to Administer the Treatment?: number analyzed (Participants) | 79 | 77
  Cycle 5. How Long Did it Take to Administer the Treatment? | 8.0 [3 to 14] | 83.0 [30 to 200]
  Cycle 5. How Long Was the Patient in the Treatment Room in Total?: number analyzed (Participants) | 79 | 77
  Cycle 5. How Long Was the Patient in the Treatment Room in Total? | 33.0 [8 to 135] | 150.0 [95 to 343]
  Cycle 6. Duration of Central Venous Catheter Set Up (IV Only)?: number analyzed (Participants) | 0 | 6
  Cycle 6. Duration of Central Venous Catheter Set Up (IV Only)? |  | 10.0 [1 to 91]
  Cycle 6. Duration of Peripherally Inserted Central Catheter Set Up (IV Only)?: number analyzed (Participants) | 0 | 0
  Cycle 6. Duration of Peripheral Vein Cannulation Set Up (IV Only)?: number analyzed (Participants) | 0 | 43
  Cycle 6. Duration of Peripheral Vein Cannulation Set Up (IV Only)? |  | 5.0 [1 to 60]
  Cycle 6. How Long Did it Take to Administer the Treatment?: number analyzed (Participants) | 79 | 80
  Cycle 6. How Long Did it Take to Administer the Treatment? | 7.0 [3 to 11] | 60.0 [5 to 275]
  Cycle 6. How Long Was the Patient in the Treatment Room in Total?: number analyzed (Participants) | 79 | 80
  Cycle 6. How Long Was the Patient in the Treatment Room in Total? | 35.0 [10 to 150] | 130.0 [45 to 330]

11. Secondary Outcome: Percentage of Healthcare Professionals (HCPs) by Their Responses on Perception of Impact of PH FDC SC on Clinical Management and Clinical Efficiency, Question 2 of the HCPQ - Treatment Room
Description: HCPs who administered study treatment responded at Cycle 6 of the Treatment Cross-Over Period to the following HCPQ-Treatment Room Question 2: "If all P+H IV infusions are switched to FDC SC injections, please indicate how strongly you agree or disagree with each of the following statements: a) Patients will be moved outside of infusion unit to receive FDC SC; b) FDC SC route will allow more flexible scheduling; c) More patients will be treated in the infusion unit; d) Waiting list for any P+H IV treatment at the infusion unit will be reduced; e) Staff resources will be redistributed to other departments of the hospital; f) There will still be sufficient interaction time between HCPs and patients; g) Staff will spend more time for further education/development; h) Staff will dedicate more time attending to administrative tasks for Perjeta-Herceptin patients; i) Patients will spend less time in the care unit; j) Administration by FDC SC injection is preferred by patients."
Time Frame: Day 1 of Cycle 6 (each cycle is 21 days)
Population: The number analyzed includes healthcare professionals (HCPs) who completed any part of the survey at treatment Cycle 6.
Measure: Number; unit: Percentage of HCPs
Groups:
- All Healthcare Professionals: This analysis set includes all healthcare professionals who treated participants from Arms A and B and completed the HCPQ questionnaire, which was administered at the last treatment cycle in the Treatment Cross-Over Period of the study. During the Treatment Cross-Over Period of the study, all participants received their first 6 cycles of treatment in accordance with the study arm to which they were randomized: Arm A) pertuzumab IV and trastuzumab IV (P+H IV) for 3 treatment cycles followed by the pertuzumab and trastuzumab fixed-dose combination for subcutaneous administration (PH FDC SC) for 3 treatment cycles (1 cycle = 21 days); or Arm B) PH FDC SC for 3 treatment cycles followed by P+H IV for 3 treatment cycles (1 cycle = 21 days). Following completion of this study period, participants chose one of the two study treatments to receive in the Treatment Continuation Period for the remaining anti-HER2 treatment cycles (18 planned cycles in total, including pre-study neoadjuvant treatment). After completing study treatment, participants entered the Follow-up Period wherein they were to be followed for 3 years from the date the last participant was randomized.
Arm/Group | All Healthcare Professionals | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 159 | 79 | 80
Percentage of HCPs
  Statement a): Strongly Disagree | 16.4 | 11.4 | 21.3
  Statement a): Disagree | 15.1 | 12.7 | 17.5
  Statement a): Neutral | 6.3 | 8.9 | 3.8
  Statement a): Agree | 21.4 | 26.6 | 16.3
  Statement a): Strongly Agree | 22.6 | 22.8 | 22.5
  Statement a): Not Applicable | 12.6 | 13.9 | 11.3
  Statement a): Answer Missing | 5.7 | 3.8 | 7.5
  Statement b): Strongly Disagree | 3.1 | 0.0 | 6.3
  Statement b): Disagree | 8.8 | 7.6 | 10.0
  Statement b): Neutral | 8.8 | 10.1 | 7.5
  Statement b): Agree | 28.3 | 29.1 | 27.5
  Statement b): Strongly Agree | 45.3 | 49.4 | 41.3
  Statement b): Not Applicable | 0.0 | 0.0 | 0.0
  Statement b): Answer Missing | 5.7 | 3.8 | 7.5
  Statement c): Strongly Disagree | 2.5 | 1.3 | 3.8
  Statement c): Disagree | 7.5 | 7.6 | 7.5
  Statement c): Neutral | 15.1 | 17.7 | 12.5
  Statement c): Agree | 30.2 | 29.1 | 31.3
  Statement c): Strongly Agree | 37.1 | 36.7 | 37.5
  Statement c): Not Applicable | 1.9 | 3.8 | 0.0
  Statement c): Answer Missing | 5.7 | 3.8 | 7.5
  Statement d): Strongly Disagree | 4.4 | 1.3 | 7.5
  Statement d): Disagree | 8.2 | 8.9 | 7.5
  Statement d): Neutral | 14.5 | 17.7 | 11.3
  Statement d): Agree | 27.7 | 29.1 | 26.3
  Statement d): Strongly Agree | 35.2 | 36.7 | 33.8
  Statement d): Not Applicable | 3.8 | 2.5 | 5.0
  Statement d): Answer Missing | 6.3 | 3.8 | 8.8
  Statement e): Strongly Disagree | 12.6 | 15.2 | 10.0
  Statement e): Disagree | 19.5 | 16.5 | 22.5
  Statement e): Neutral | 20.1 | 17.7 | 22.5
  Statement e): Agree | 15.1 | 19.0 | 11.3
  Statement e): Strongly Agree | 19.5 | 20.3 | 18.8
  Statement e): Not Applicable | 6.9 | 7.6 | 6.3
  Statement e): Answer Missing | 6.3 | 3.8 | 8.8
  Statement f): Strongly Disagree | 1.9 | 0.0 | 3.8
  Statement f): Disagree | 5.0 | 6.3 | 3.8
  Statement f): Neutral | 15.7 | 15.2 | 16.3
  Statement f): Agree | 32.1 | 31.6 | 32.5
  Statement f): Strongly Agree | 39.0 | 43.0 | 35.0
  Statement f): Not Applicable | 0.0 | 0.0 | 0.0
  Statement f): Answer Missing | 6.3 | 3.8 | 8.8
  Statement g): Strongly Disagree | 2.5 | 0.0 | 5.0
  Statement g): Disagree | 9.4 | 7.6 | 11.3
  Statement g): Neutral | 27.7 | 31.6 | 23.8
  Statement g): Agree | 21.4 | 20.3 | 22.5
  Statement g): Strongly Agree | 31.4 | 35.4 | 27.5
  Statement g): Not Applicable | 1.9 | 1.3 | 2.5
  Statement g): Answer Missing | 5.7 | 3.8 | 7.5
  Statement h): Strongly Disagree | 3.1 | 1.3 | 5.0
  Statement h): Disagree | 13.8 | 11.4 | 16.3
  Statement h): Neutral | 24.5 | 25.3 | 23.8
  Statement h): Agree | 20.1 | 24.1 | 16.3
  Statement h): Strongly Agree | 30.2 | 32.9 | 27.5
  Statement h): Not Applicable | 2.5 | 1.3 | 3.8
  Statement h): Answer Missing | 5.7 | 3.8 | 7.5
  Statement i): Strongly Disagree | 0.0 | 0.0 | 0.0
  Statement i): Disagree | 5.0 | 6.3 | 3.8
  Statement i): Neutral | 3.1 | 1.3 | 5.0
  Statement i): Agree | 25.2 | 27.8 | 22.5
  Statement i): Strongly Agree | 60.4 | 60.8 | 60.0
  Statement i): Not Applicable | 0.0 | 0.0 | 0.0
  Statement i): Answer Missing | 6.3 | 3.8 | 8.8
  Statement j): Strongly Disagree | 0.0 | 0.0 | 0.0
  Statement j): Disagree | 5.0 | 8.9 | 1.3
  Statement j): Neutral | 12.6 | 10.1 | 15.0
  Statement j): Agree | 24.5 | 22.8 | 26.3
  Statement j): Strongly Agree | 50.3 | 53.2 | 47.5
  Statement j): Not Applicable | 1.3 | 1.3 | 1.3
  Statement j): Answer Missing | 6.3 | 3.8 | 8.8

12. Secondary Outcome: Percentage of Healthcare Professionals (HCPs) by Their Responses on Perception of Time/Resource Use and Convenience of Each Study Regimen, Questions 3 to 7 of the HCPQ - Treatment Room
Description: Healthcare professionals (HCPs) who administered study treatment responded at Cycle 6 of the Treatment Cross-Over Period to the following HCPQ-Treatment Room Questions 3 to 7: "Looking back over the Perjeta-Herceptin treatment sessions, please indicate based on your opinion which administration method: Q3. Which Method Was Most Convenient for the Patient? Q4. Which Method Was Best for Optimizing Patient Care in Your Centre? Q5. Which Method Took the Least Time from Start to Finish of Administration? Q6. Which Method Required the Least Resource Use for Administration? Q7. Which Method Was Preferred by Patients?" The four available response options were: P+H IV, FDC SC, No Difference, and Unsure.
Time Frame: Day 1 of Cycle 6 (each cycle is 21 days)
Population: The number analyzed includes HCPs who completed any part of the survey at treatment Cycle 6.
Measure: Number; unit: Percentage of HCPs
Arm/Group | All Healthcare Professionals | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 159 | 79 | 80
Percentage of HCPs
  Q3. Answer: FDC SC | 86.8 | 88.6 | 85.0
  Q3. Answer: P+H IV | 3.8 | 6.3 | 1.3
  Q3. Answer: No Difference | 3.8 | 2.5 | 5.0
  Q3. Answer: Unsure | 3.8 | 0.0 | 7.5
  Q3. Answer: Missing | 1.9 | 2.5 | 1.3
  Q4. Answer: FDC SC | 79.2 | 79.7 | 78.8
  Q4. Answer: P+H IV | 2.5 | 3.8 | 1.3
  Q4. Answer: No Difference | 12.6 | 12.7 | 12.5
  Q4. Answer: Unsure | 3.8 | 1.3 | 6.3
  Q4. Answer: Missing | 1.9 | 2.5 | 1.3
  Q5. Answer: FDC SC | 95.6 | 94.9 | 96.3
  Q5. Answer: P+H IV | 0.0 | 0.0 | 0.0
  Q5. Answer: No Difference | 2.5 | 2.5 | 2.5
  Q5. Answer: Unsure | 0.0 | 0.0 | 0.0
  Q5. Answer: Missing | 1.9 | 2.5 | 1.3
  Q6. Answer: FDC SC | 86.2 | 83.5 | 88.8
  Q6. Answer: P+H IV | 0.6 | 0.0 | 1.3
  Q6. Answer: No Difference | 11.3 | 13.9 | 8.8
  Q6. Answer: Unsure | 0.0 | 0.0 | 0.0
  Q6. Answer: Missing | 1.9 | 2.5 | 1.3
  Q7. Answer: FDC SC | 77.4 | 77.2 | 77.5
  Q7. Answer: P+H IV | 6.3 | 7.6 | 5.0
  Q7. Answer: No Difference | 2.5 | 2.5 | 2.5
  Q7. Answer: Unsure | 11.9 | 10.1 | 13.8
  Q7. Answer: Missing | 1.9 | 2.5 | 1.3

13. Secondary Outcome: Percentage of Healthcare Professionals (HCPs) by Their Responses to Question 8 of the HCPQ - Treatment Room
Description: Healthcare professionals (HCPs) who administered study treatment responded at Cycle 6 of the Treatment Cross-Over Period to the following HCPQ-Treatment Room Question 8: "How frequently would you offer or recommend FDC SC administration to your patients in the future?" The three available response options were: Always, Sometimes, and Never.
Time Frame: Day 1 of Cycle 6 (each cycle is 21 days)
Population: The number analyzed includes HCPs who completed any part of the survey at treatment Cycle 6.
Measure: Number; unit: Percentage of HCPs
Arm/Group | All Healthcare Professionals | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 159 | 79 | 80
Percentage of HCPs
  Always | 67.3 | 69.6 | 65.0
  Sometimes | 30.2 | 26.6 | 33.8
  Never | 0.6 | 1.3 | 0.0
  Missing | 1.9 | 2.5 | 1.3

14. Secondary Outcome: Duration of Treatment Preparation According to Healthcare Professionals' Responses on Perception of Time by Treatment Cycle, Question 1 of the HCPQ - Drug Preparation Room
Description: The Healthcare Professional Questionnaire (HCPQ)-Drug Preparation Room Question 1 was completed at each treatment cycle of the Treatment Cross-Over Period by the healthcare professionals (HCPs) within the pharmacy/drug preparation area where pertuzumab IV and trastuzumab IV and pertuzumab and trastuzumab FDC SC were prepared and dispensed for treating the study's participants. HCPs responded to the following question: "How long (in minutes) did it take to prepare the treatment for use?"
Time Frame: Day 1 of Cycles 1-6 (each cycle is 21 days)
Population: The number analyzed includes healthcare professionals (HCPs) who completed question 1 of the survey per treatment cycle.
Measure: Median (Full Range); unit: minutes
Arm/Group | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 80 | 80
minutes
  Cycle 1: number analyzed (Participants) | 80 | 79
  Cycle 1 | 20.0 [3 to 60] | 5.0 [1 to 50]
  Cycle 2: number analyzed (Participants) | 79 | 80
  Cycle 2 | 20.0 [3 to 60] | 5.0 [1 to 30]
  Cycle 3: number analyzed (Participants) | 80 | 79
  Cycle 3 | 17.5 [3 to 90] | 5.0 [1 to 40]
  Cycle 4 | 5.0 [1 to 30] | 15.0 [3 to 49]
  Cycle 5: number analyzed (Participants) | 80 | 79
  Cycle 5 | 5.0 [1 to 35] | 15.0 [3 to 50]
  Cycle 6: number analyzed (Participants) | 80 | 78
  Cycle 6 | 5.0 [1 to 40] | 15.0 [3 to 50]

15. Secondary Outcome: Percentage of Healthcare Professionals (HCPs) by Their Responses on Perception of Impact of PH FDC SC on Clinical Management and Clinical Efficiency, Question 2 of the HCPQ - Drug Preparation Room
Description: Healthcare professionals (HCPs) who prepared study treatment within the pharmacy/drug preparation area responded at Cycle 6 of the Treatment Cross-Over Period to the following HCPQ-Drug Preparation Room Question 2: "If all P+H IV infusions are switched to FDC SC injections, please indicate how strongly you agree or disagree with each of the following statements: a) Staff will have increased availability for other tasks in the pharmacy; b) Administrative procedures around FDC SC will require less time; c) FDC SC formulations will provide more flexibility for staff in managing their workload; d) Due to ready-to-use FDC SC formulations, potential dosing errors will be avoided; e) Due to ready-to-use FDC SC formulations, there will be less drug wastage; f) Without having to reconstitute the drug, less storage space for FDC SC related supplies will be required in the pharmacy; g) Preparation procedures and associated time staff time commitment will be reduced."
Time Frame: Day 1 of Cycle 6 (each cycle is 21 days)
Population: The number analyzed includes healthcare professionals (HCPs) who completed any part of the survey at treatment Cycle 6.
Measure: Number; unit: Percentage of HCPs
Arm/Group | All Healthcare Professionals | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 160 | 80 | 80
Percentage of HCPs
  Statement a): Strongly Disagree | 1.3 | 1.3 | 1.3
  Statement a): Disagree | 0.6 | 1.3 | 0.0
  Statement a): Neutral | 7.5 | 8.8 | 6.3
  Statement a): Agree | 28.8 | 28.8 | 28.8
  Statement a): Strongly Agree | 50.6 | 52.5 | 48.8
  Statement a): Not Applicable | 2.5 | 3.8 | 1.3
  Statement a): Answer Missing | 8.8 | 3.8 | 13.8
  Statement b): Strongly Disagree | 5.6 | 8.8 | 2.5
  Statement b): Disagree | 3.8 | 3.8 | 3.8
  Statement b): Neutral | 14.4 | 16.3 | 12.5
  Statement b): Agree | 18.1 | 17.5 | 18.8
  Statement b): Strongly Agree | 46.3 | 46.3 | 46.3
  Statement b): Not Applicable | 2.5 | 2.5 | 2.5
  Statement b): Answer Missing | 9.4 | 5.0 | 13.8
  Statement c): Strongly Disagree | 0.6 | 0.0 | 1.3
  Statement c): Disagree | 0.6 | 0.0 | 1.3
  Statement c): Neutral | 13.1 | 15.0 | 11.3
  Statement c): Agree | 26.3 | 28.8 | 23.8
  Statement c): Strongly Agree | 48.8 | 50.0 | 47.5
  Statement c): Not Applicable | 1.3 | 1.3 | 1.3
  Statement c): Answer Missing | 9.4 | 5.0 | 13.8
  Statement d): Strongly Disagree | 1.3 | 1.3 | 1.3
  Statement d): Disagree | 3.8 | 1.3 | 6.3
  Statement d): Neutral | 5.6 | 5.0 | 6.3
  Statement d): Agree | 23.1 | 26.3 | 20.0
  Statement d): Strongly Agree | 56.3 | 60.0 | 52.5
  Statement d): Not Applicable | 1.3 | 1.3 | 1.3
  Statement d): Answer Missing | 8.8 | 5.0 | 12.5
  Statement e): Strongly Disagree | 1.3 | 1.3 | 1.3
  Statement e): Disagree | 1.9 | 1.3 | 2.5
  Statement e): Neutral | 8.8 | 11.3 | 6.3
  Statement e): Agree | 21.9 | 21.3 | 22.5
  Statement e): Strongly Agree | 55.0 | 58.8 | 51.3
  Statement e): Not Applicable | 1.9 | 1.3 | 2.5
  Statement e): Answer Missing | 9.4 | 5.0 | 13.8
  Statement f): Strongly Disagree | 0.6 | 0.0 | 1.3
  Statement f): Disagree | 4.4 | 3.8 | 5.0
  Statement f): Neutral | 11.9 | 16.3 | 7.5
  Statement f): Agree | 24.4 | 20.0 | 28.8
  Statement f): Strongly Agree | 48.1 | 53.8 | 42.5
  Statement f): Not Applicable | 1.3 | 1.3 | 1.3
  Statement f): Answer Missing | 9.4 | 5.0 | 13.8
  Statement g): Strongly Disagree | 0.6 | 0.0 | 1.3
  Statement g): Disagree | 0.0 | 0.0 | 0.0
  Statement g): Neutral | 6.9 | 8.8 | 5.0
  Statement g): Agree | 31.3 | 30.0 | 32.5
  Statement g): Strongly Agree | 48.8 | 52.5 | 45.0
  Statement g): Not Applicable | 3.1 | 3.8 | 2.5
  Statement g): Answer Missing | 9.4 | 5.0 | 13.8

16. Secondary Outcome: Percentage of Healthcare Professionals (HCPs) by Their Responses on Perception of Time/Resource Use of Each Study Regimen, Questions 3 and 4 of the HCPQ - Drug Preparation Room
Description: Healthcare professionals (HCPs) who prepared study treatment within the pharmacy/drug preparation area responded at Cycle 6 of the Treatment Cross-Over Period to the following HCPQ-Drug Preparation Room Questions 3 and 4: "Looking back over the Perjeta-Herceptin treatment sessions, please indicate based on your opinion which administration method: Q3. Was quickest from start to end of preparation to finish of administration (excluding observation period)?; Q4. Required less resource use for preparation and administration, for example nursing time, facility costs, equipment etc?" The three available response options were: P+H IV, FDC SC, and No Difference.
Time Frame: Day 1 of Cycle 6 (each cycle is 21 days)
Population: The number analyzed includes healthcare professionals (HCPs) who completed any part of the survey at treatment Cycle 6.
Measure: Number; unit: Percentage of HCPs
Arm/Group | All Healthcare Professionals | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 160 | 80 | 80
Percentage of HCPs
  Q3. Answer: FDC SC | 87.5 | 92.5 | 82.5
  Q3. Answer: P+H IV | 0.6 | 0.0 | 1.3
  Q3. Answer: No Difference | 1.3 | 1.3 | 1.3
  Q3. Answer: Missing | 10.6 | 6.3 | 15.0
  Q4. Answer: FDC SC | 86.9 | 93.8 | 80.0
  Q4. Answer: P+H IV | 0.0 | 0.0 | 0.0
  Q4. Answer: No Difference | 2.5 | 0.0 | 5.0
  Q4. Answer: Missing | 10.6 | 6.3 | 15.0

17. Secondary Outcome: Change From Baseline Over Time in Health-Related Quality of Life (HRQoL) as Assessed by the Global Health Status (GHS)/HRQoL Scale Score of the the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire 30 (EORTC QLQ-C30)
Description: The EORTC QLQ-C30 questionnaire consisted of 30 questions covering treatment-related symptoms, functioning, and GHS/HRQoL. Questions were answered by participants on a scale from 1 to 4 or 1 to 7. Raw scores were transformed to scale scores that ranged from 0 to 100 where a higher scale score indicating a higher response (i.e., on the functioning and GHS/QoL scales a higher score meant better functioning/QoL, whereas on the symptom scales a higher score meant greater [worse] symptoms). The EORTC QLQ-C30 data was scored according to the EORTC scoring manual (Fayers 2001). In the event of incomplete data, for all questionnaire subscales, if more than 50% of the constituent items are completed, a pro-rated score was to be computed consistent with the scoring manuals and published validation reports. For subscales with less than 50% of the items completed, the subscale was to be considered as missing.
Time Frame: Baseline (Day 1 of Cycle 1); Day 1 of Cycles 3, 6, and 15 (or last treatment cycle; each cycle is 21 days); 1.5, 2, and 3 years (up to 3 years)
Population: The Patient-Reported Outcome (PRO)-Evaluable Population includes all participants in the ITT population with a baseline EORTC QLQ-C30 assessment and at least one post-baseline EORTC QLQ-C30 assessment. The number analyzed at a given timepoint indicates participants with non-missing data at that timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 159 | 79 | 80
score on a scale
  Baseline (BL): Value at Visit | 74.21 (16.79) | 71.62 (17.98) | 76.77 (15.22)
  Change from BL at Cycle 3 Day 1: number analyzed (Participants) | 157 | 77 | 80
  Change from BL at Cycle 3 Day 1 | 0.27 (15.72) | 0.54 (16.63) | 0.00 (14.88)
  Change from BL at Cycle 6 Day 1: number analyzed (Participants) | 155 | 76 | 79
  Change from BL at Cycle 6 Day 1 | -0.05 (18.38) | 1.10 (20.25) | -1.16 (16.44)
  Change from BL at Cycle 15 or Last Treatment Cycle: number analyzed (Participants) | 142 | 71 | 71
  Change from BL at Cycle 15 or Last Treatment Cycle | 2.29 (17.05) | 2.82 (16.30) | 1.76 (17.87)
  Change from BL at 1.5 Years: number analyzed (Participants) | 146 | 72 | 74
  Change from BL at 1.5 Years | 6.79 (19.38) | 7.18 (21.73) | 6.42 (16.92)
  Change from BL at 2 Years: number analyzed (Participants) | 146 | 73 | 73
  Change from BL at 2 Years | 5.14 (18.45) | 6.16 (19.45) | 4.11 (17.46)
  Change from BL at 3 Years: number analyzed (Participants) | 133 | 68 | 65
  Change from BL at 3 Years | 6.89 (18.45) | 7.23 (16.85) | 6.54 (20.12)

18. Secondary Outcome: Change From Baseline Over Time in the Physical Functioning Scale Score of the EORTC QLQ-C30
Description: as for outcome 17
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 159 | 79 | 80
score on a scale
  Baseline (BL): Value at Visit | 86.16 (14.48) | 84.22 (14.91) | 88.08 (13.86)
  Change from BL at Cycle 3 Day 1 | 0.67 (12.08) | 1.77 (12.97) | -0.42 (11.09)
  Change from BL at Cycle 6 Day 1: number analyzed (Participants) | 155 | 76 | 79
  Change from BL at Cycle 6 Day 1 | 1.20 (14.46) | 1.93 (16.61) | 0.51 (12.11)
  Change from BL at Cycle 15 or Last Treatment Cycle: number analyzed (Participants) | 142 | 71 | 71
  Change from BL at Cycle 15 or Last Treatment Cycle | 2.54 (15.79) | 3.85 (13.65) | 1.22 (17.69)
  Change from BL at 1.5 Years: number analyzed (Participants) | 146 | 72 | 74
  Change from BL at 1.5 Years | 4.74 (15.71) | 5.44 (17.29) | 4.05 (14.08)
  Change from BL at 2 Years: number analyzed (Participants) | 146 | 73 | 73
  Change from BL at 2 Years | 3.97 (16.32) | 4.38 (18.57) | 3.56 (13.84)
  Change from BL at 3 Years: number analyzed (Participants) | 133 | 68 | 65
  Change from BL at 3 Years | 2.51 (14.67) | 3.33 (13.99) | 1.64 (15.41)

19. Secondary Outcome: Change From Baseline Over Time in the Role Functioning Scale Score of the EORTC QLQ-C30
Description: as for outcome 17
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 159 | 79 | 80
score on a scale
  Baseline (BL): Value at Visit | 78.30 (25.76) | 79.54 (25.45) | 77.08 (26.17)
  Change from BL at Cycle 3 Day 1 | 6.71 (25.37) | 3.80 (24.01) | 9.58 (26.49)
  Change from BL at Cycle 6 Day 1: number analyzed (Participants) | 155 | 76 | 79
  Change from BL at Cycle 6 Day 1 | 7.42 (26.12) | 6.36 (24.03) | 8.44 (28.10)
  Change from BL at Cycle 15 or Last Treatment Cycle: number analyzed (Participants) | 142 | 71 | 71
  Change from BL at Cycle 15 or Last Treatment Cycle | 9.62 (29.60) | 6.81 (24.00) | 12.44 (34.24)
  Change from BL at 1.5 Years: number analyzed (Participants) | 146 | 72 | 74
  Change from BL at 1.5 Years | 13.24 (30.00) | 9.49 (29.31) | 16.89 (30.41)
  Change from BL at 2 Years: number analyzed (Participants) | 146 | 73 | 73
  Change from BL at 2 Years | 11.30 (30.07) | 11.64 (29.22) | 10.96 (31.08)
  Change from BL at 3 Years: number analyzed (Participants) | 133 | 68 | 65
  Change from BL at 3 Years | 10.40 (29.13) | 8.09 (26.78) | 12.82 (31.43)

20. Secondary Outcome: Change From Baseline Over Time in the Emotional Functioning Scale Score of the EORTC QLQ-C30
Description: as for outcome 17
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 159 | 79 | 80
score on a scale
  Baseline (BL): Value at Visit | 82.08 (17.72) | 82.07 (16.99) | 82.08 (18.52)
  Change from BL at Cycle 3 Day 1: number analyzed (Participants) | 158 | 78 | 80
  Change from BL at Cycle 3 Day 1 | 0.05 (15.92) | -1.28 (15.26) | 1.35 (16.53)
  Change from BL at Cycle 6 Day 1: number analyzed (Participants) | 155 | 76 | 79
  Change from BL at Cycle 6 Day 1 | 0.32 (18.70) | 0.99 (20.04) | -0.32 (17.42)
  Change from BL at Cycle 15 or Last Treatment Cycle: number analyzed (Participants) | 142 | 71 | 71
  Change from BL at Cycle 15 or Last Treatment Cycle | 0.65 (19.60) | -1.17 (15.77) | 2.46 (22.77)
  Change from BL at 1.5 Years: number analyzed (Participants) | 146 | 72 | 74
  Change from BL at 1.5 Years | 2.45 (22.47) | 0.93 (23.05) | 3.94 (21.95)
  Change from BL at 2 Years: number analyzed (Participants) | 146 | 73 | 73
  Change from BL at 2 Years | 1.86 (23.78) | 2.74 (21.61) | 0.99 (25.89)
  Change from BL at 3 Years: number analyzed (Participants) | 133 | 68 | 65
  Change from BL at 3 Years | 2.38 (23.78) | 3.55 (21.08) | 1.15 (26.43)

21. Secondary Outcome: Change From Baseline Over Time in the Cognitive Functioning Scale Score of the EORTC QLQ-C30
Description: as for outcome 17
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 159 | 79 | 80
score on a scale
  Baseline (BL): Value at Visit | 85.22 (18.37) | 85.86 (17.92) | 84.58 (18.90)
  Change from BL at Cycle 3 Day 1: number analyzed (Participants) | 158 | 78 | 80
  Change from BL at Cycle 3 Day 1 | -0.95 (19.21) | -0.64 (17.08) | -1.25 (21.18)
  Change from BL at Cycle 6 Day 1: number analyzed (Participants) | 155 | 76 | 79
  Change from BL at Cycle 6 Day 1 | -2.47 (20.44) | -3.29 (18.86) | -1.69 (21.94)
  Change from BL at Cycle 15 or Last Treatment Cycle: number analyzed (Participants) | 142 | 71 | 71
  Change from BL at Cycle 15 or Last Treatment Cycle | -4.69 (22.58) | -7.75 (21.79) | -1.64 (23.09)
  Change from BL at 1.5 Years: number analyzed (Participants) | 146 | 72 | 74
  Change from BL at 1.5 Years | -1.94 (21.31) | -3.47 (20.16) | -0.45 (22.41)
  Change from BL at 2 Years: number analyzed (Participants) | 146 | 73 | 73
  Change from BL at 2 Years | -1.03 (21.10) | -2.51 (20.54) | 0.46 (21.69)
  Change from BL at 3 Years: number analyzed (Participants) | 133 | 68 | 65
  Change from BL at 3 Years | -3.01 (23.64) | -2.45 (20.42) | -3.59 (26.76)

22. Secondary Outcome: Change From Baseline Over Time in the Social Functioning Scale Score of the EORTC QLQ-C30
Description: as for outcome 17
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 158 | 78 | 80
score on a scale
  Baseline (BL): Value at Visit | 79.01 (21.79) | 77.99 (22.39) | 80.00 (21.28)
  Change from BL at Cycle 3 Day 1: number analyzed (Participants) | 157 | 77 | 80
  Change from BL at Cycle 3 Day 1 | 6.26 (22.60) | 5.41 (24.40) | 7.08 (20.84)
  Change from BL at Cycle 6 Day 1: number analyzed (Participants) | 154 | 75 | 79
  Change from BL at Cycle 6 Day 1 | 4.44 (22.87) | 6.44 (25.39) | 2.53 (20.16)
  Change from BL at Cycle 15 or Last Treatment Cycle: number analyzed (Participants) | 141 | 70 | 71
  Change from BL at Cycle 15 or Last Treatment Cycle | 7.80 (23.87) | 9.05 (23.86) | 6.57 (23.98)
  Change from BL at 1.5 Years: number analyzed (Participants) | 145 | 71 | 74
  Change from BL at 1.5 Years | 12.41 (24.20) | 12.21 (29.41) | 12.61 (18.05)
  Change from BL at 2 Years: number analyzed (Participants) | 145 | 72 | 73
  Change from BL at 2 Years | 13.68 (24.19) | 15.28 (25.29) | 12.10 (23.12)
  Change from BL at 3 Years: number analyzed (Participants) | 132 | 67 | 65
  Change from BL at 3 Years | 12.63 (24.46) | 11.94 (25.76) | 13.33 (23.24)

23. Secondary Outcome: Change From Baseline Over Time in the Fatigue Scale Score of the EORTC QLQ-C30
Description: as for outcome 17
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 159 | 79 | 80
score on a scale
  Baseline (BL): Value at Visit | 22.01 (18.90) | 24.47 (19.28) | 19.58 (18.31)
  Change from BL at Cycle 3 Day 1 | 1.29 (16.35) | -0.14 (17.66) | 2.71 (14.92)
  Change from BL at Cycle 6 Day 1: number analyzed (Participants) | 155 | 76 | 79
  Change from BL at Cycle 6 Day 1 | 0.50 (19.22) | -3.22 (17.85) | 4.08 (19.91)
  Change from BL at Cycle 15 or Last Treatment Cycle: number analyzed (Participants) | 142 | 71 | 71
  Change from BL at Cycle 15 or Last Treatment Cycle | -2.11 (21.46) | -3.44 (18.36) | -0.78 (24.22)
  Change from BL at 1.5 Years: number analyzed (Participants) | 146 | 72 | 74
  Change from BL at 1.5 Years | -7.76 (19.59) | -9.26 (20.43) | -6.31 (18.76)
  Change from BL at 2 Years: number analyzed (Participants) | 146 | 73 | 73
  Change from BL at 2 Years | -5.25 (24.49) | -6.54 (25.51) | -3.96 (23.52)
  Change from BL at 3 Years: number analyzed (Participants) | 133 | 68 | 65
  Change from BL at 3 Years | -5.43 (22.58) | -7.68 (21.66) | -3.08 (23.45)

24. Secondary Outcome: Change From Baseline Over Time in the Nausea and Vomiting Scale Score of the EORTC QLQ-C30
Description: as for outcome 17
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 159 | 79 | 80
score on a scale
  Baseline (BL): Value at Visit | 2.73 (8.57) | 2.11 (7.24) | 3.33 (9.71)
  Change from BL at Cycle 3 Day 1 | 0.84 (10.74) | 0.21 (9.80) | 1.46 (11.62)
  Change from BL at Cycle 6 Day 1: number analyzed (Participants) | 155 | 76 | 79
  Change from BL at Cycle 6 Day 1 | 0.75 (11.61) | 1.54 (11.92) | 0.00 (11.32)
  Change from BL at Cycle 15 or Last Treatment Cycle: number analyzed (Participants) | 142 | 71 | 71
  Change from BL at Cycle 15 or Last Treatment Cycle | 1.17 (11.34) | 1.88 (12.13) | 0.47 (10.53)
  Change from BL at 1.5 Years: number analyzed (Participants) | 146 | 72 | 74
  Change from BL at 1.5 Years | -0.23 (11.41) | 0.46 (11.18) | -0.90 (11.67)
  Change from BL at 2 Years: number analyzed (Participants) | 146 | 73 | 73
  Change from BL at 2 Years | -0.68 (11.05) | -0.23 (11.28) | -1.14 (10.88)
  Change from BL at 3 Years: number analyzed (Participants) | 133 | 68 | 65
  Change from BL at 3 Years | -0.75 (10.83) | -1.23 (9.69) | -0.26 (11.97)

25. Secondary Outcome: Change From Baseline Over Time in the Pain Scale Score of the EORTC QLQ-C30
Description: as for outcome 17
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 159 | 79 | 80
score on a scale
  Baseline (BL): Value at Visit | 16.04 (22.26) | 17.72 (24.94) | 14.38 (19.26)
  Change from BL at Cycle 3 Day 1 | 0.21 (25.02) | 0.00 (27.86) | 0.42 (22.02)
  Change from BL at Cycle 6 Day 1: number analyzed (Participants) | 155 | 76 | 79
  Change from BL at Cycle 6 Day 1 | 0.43 (23.34) | -2.41 (25.92) | 3.16 (20.34)
  Change from BL at Cycle 15 or Last Treatment Cycle: number analyzed (Participants) | 142 | 71 | 71
  Change from BL at Cycle 15 or Last Treatment Cycle | -1.17 (25.85) | -2.82 (25.04) | 0.47 (26.72)
  Change from BL at 1.5 Years: number analyzed (Participants) | 146 | 72 | 74
  Change from BL at 1.5 Years | -1.26 (28.84) | -1.62 (33.47) | -0.90 (23.71)
  Change from BL at 2 Years: number analyzed (Participants) | 146 | 73 | 73
  Change from BL at 2 Years | -3.08 (26.91) | -1.83 (30.25) | -4.34 (23.25)
  Change from BL at 3 Years: number analyzed (Participants) | 133 | 68 | 65
  Change from BL at 3 Years | -2.13 (28.23) | -1.72 (26.88) | -2.56 (29.79)

26. Secondary Outcome: Change From Baseline Over Time in the Dyspnoea Scale Score of the EORTC QLQ-C30
Description: as for outcome 17
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 159 | 79 | 80
score on a scale
  Baseline (BL): Value at Visit | 5.87 (15.25) | 6.75 (15.45) | 5.00 (15.09)
  Change from BL at Cycle 3 Day 1 | 0.63 (13.24) | -0.42 (14.61) | 1.67 (11.74)
  Change from BL at Cycle 6 Day 1: number analyzed (Participants) | 155 | 76 | 79
  Change from BL at Cycle 6 Day 1 | 3.01 (15.83) | 1.32 (15.81) | 4.64 (15.77)
  Change from BL at Cycle 15 or Last Treatment Cycle: number analyzed (Participants) | 142 | 71 | 71
  Change from BL at Cycle 15 or Last Treatment Cycle | 1.88 (17.65) | 1.41 (19.05) | 2.35 (16.26)
  Change from BL at 1.5 Years: number analyzed (Participants) | 146 | 72 | 74
  Change from BL at 1.5 Years | 0.68 (13.82) | -0.46 (10.46) | 1.80 (16.45)
  Change from BL at 2 Years: number analyzed (Participants) | 146 | 73 | 73
  Change from BL at 2 Years | 1.83 (14.00) | 1.83 (16.56) | 1.83 (10.96)
  Change from BL at 3 Years: number analyzed (Participants) | 133 | 68 | 65
  Change from BL at 3 Years | 1.50 (14.13) | 1.47 (13.42) | 1.54 (14.94)

27. Secondary Outcome: Change From Baseline Over Time in the Insomnia Scale Score of the EORTC QLQ-C30
Description: as for outcome 17
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 159 | 79 | 80
score on a scale
  Baseline (BL): Value at Visit | 22.22 (25.34) | 21.94 (24.97) | 22.50 (25.86)
  Change from BL at Cycle 3 Day 1 | 1.26 (27.01) | 2.95 (26.25) | -0.42 (27.81)
  Change from BL at Cycle 6 Day 1: number analyzed (Participants) | 155 | 76 | 79
  Change from BL at Cycle 6 Day 1 | 1.72 (29.86) | 5.26 (29.34) | -1.69 (30.15)
  Change from BL at Cycle 15 or Last Treatment Cycle: number analyzed (Participants) | 142 | 71 | 71
  Change from BL at Cycle 15 or Last Treatment Cycle | -0.94 (31.75) | 3.76 (32.15) | -5.63 (30.85)
  Change from BL at 1.5 Years: number analyzed (Participants) | 146 | 72 | 74
  Change from BL at 1.5 Years | -0.23 (30.95) | 1.85 (30.07) | -2.25 (31.85)
  Change from BL at 2 Years: number analyzed (Participants) | 146 | 73 | 73
  Change from BL at 2 Years | 2.97 (33.89) | 6.85 (35.56) | -0.91 (31.90)
  Change from BL at 3 Years: number analyzed (Participants) | 133 | 68 | 65
  Change from BL at 3 Years | 0.00 (34.08) | 1.47 (33.79) | -1.54 (34.58)

28. Secondary Outcome: Change From Baseline Over Time in the Appetite Loss Scale Score of the EORTC QLQ-C30
Description: as for outcome 17
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 159 | 79 | 80
score on a scale
  Baseline (BL): Value at Visit | 10.06 (19.40) | 8.44 (14.59) | 11.67 (23.18)
  Change from BL at Cycle 3 Day 1 | 0.21 (21.38) | 3.38 (23.02) | -2.92 (19.26)
  Change from BL at Cycle 6 Day 1: number analyzed (Participants) | 155 | 76 | 79
  Change from BL at Cycle 6 Day 1 | -0.86 (18.20) | 0.00 (18.86) | -1.69 (17.62)
  Change from BL at Cycle 15 or Last Treatment Cycle: number analyzed (Participants) | 142 | 71 | 71
  Change from BL at Cycle 15 or Last Treatment Cycle | -5.40 (20.49) | -4.69 (17.18) | -6.10 (23.44)
  Change from BL at 1.5 Years: number analyzed (Participants) | 146 | 72 | 74
  Change from BL at 1.5 Years | -6.16 (19.96) | -4.63 (20.41) | -7.66 (19.54)
  Change from BL at 2 Years: number analyzed (Participants) | 146 | 73 | 73
  Change from BL at 2 Years | -4.34 (18.47) | -5.48 (15.73) | -3.20 (20.91)
  Change from BL at 3 Years: number analyzed (Participants) | 133 | 68 | 65
  Change from BL at 3 Years | -6.02 (19.61) | -5.39 (15.89) | -6.67 (22.97)

29. Secondary Outcome: Change From Baseline Over Time in the Constipation Scale Score of the EORTC QLQ-C30
Description: as for outcome 17
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 159 | 79 | 80
score on a scale
  Baseline (BL): Value at Visit | 9.01 (19.37) | 8.44 (16.42) | 9.58 (21.99)
  Change from BL at Cycle 3 Day 1 | -1.68 (16.69) | 0.00 (15.10) | -3.33 (18.06)
  Change from BL at Cycle 6 Day 1: number analyzed (Participants) | 155 | 76 | 79
  Change from BL at Cycle 6 Day 1 | -0.86 (19.35) | 0.88 (20.35) | -2.53 (18.31)
  Change from BL at Cycle 15 or Last Treatment Cycle: number analyzed (Participants) | 142 | 71 | 71
  Change from BL at Cycle 15 or Last Treatment Cycle | -0.70 (21.18) | 0.00 (20.31) | -1.41 (22.14)
  Change from BL at 1.5 Years: number analyzed (Participants) | 146 | 72 | 74
  Change from BL at 1.5 Years | 0.23 (23.97) | 0.00 (17.69) | 0.45 (28.93)
  Change from BL at 2 Years: number analyzed (Participants) | 146 | 73 | 73
  Change from BL at 2 Years | 1.60 (26.93) | 5.94 (26.26) | -2.74 (27.08)
  Change from BL at 3 Years: number analyzed (Participants) | 133 | 68 | 65
  Change from BL at 3 Years | 1.50 (23.52) | 0.49 (20.36) | 2.56 (26.55)

30. Secondary Outcome: Change From Baseline Over Time in the Diarrhoea Scale Score of the EORTC QLQ-C30
Description: as for outcome 17
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 159 | 79 | 80
score on a scale
  Baseline (BL): Value at Visit | 10.48 (21.59) | 12.24 (22.76) | 8.75 (20.36)
  Change from BL at Cycle 3 Day 1: number analyzed (Participants) | 158 | 78 | 80
  Change from BL at Cycle 3 Day 1 | 7.17 (27.22) | 4.70 (25.04) | 9.58 (29.14)
  Change from BL at Cycle 6 Day 1: number analyzed (Participants) | 155 | 76 | 79
  Change from BL at Cycle 6 Day 1 | 4.95 (24.26) | 4.39 (23.31) | 5.49 (25.28)
  Change from BL at Cycle 15 or Last Treatment Cycle: number analyzed (Participants) | 142 | 71 | 71
  Change from BL at Cycle 15 or Last Treatment Cycle | 2.58 (26.06) | 2.82 (25.66) | 2.35 (26.62)
  Change from BL at 1.5 Years: number analyzed (Participants) | 146 | 72 | 74
  Change from BL at 1.5 Years | -6.39 (22.25) | -8.33 (23.57) | -4.50 (20.88)
  Change from BL at 2 Years: number analyzed (Participants) | 146 | 73 | 73
  Change from BL at 2 Years | -6.85 (23.79) | -8.22 (26.52) | -5.48 (20.80)
  Change from BL at 3 Years: number analyzed (Participants) | 133 | 68 | 65
  Change from BL at 3 Years | -7.52 (23.79) | -9.80 (25.79) | -5.13 (21.43)

31. Secondary Outcome: Change From Baseline Over Time in the Financial Difficulties Scale Score of the EORTC QLQ-C30
Description: as for outcome 17
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 159 | 79 | 80
score on a scale
  Baseline (BL): Value at Visit | 22.85 (27.59) | 23.63 (27.30) | 22.08 (28.04)
  Change from BL at Cycle 3 Day 1: number analyzed (Participants) | 158 | 78 | 80
  Change from BL at Cycle 3 Day 1 | -2.95 (22.38) | -2.99 (20.23) | -2.92 (24.42)
  Change from BL at Cycle 6 Day 1: number analyzed (Participants) | 155 | 76 | 79
  Change from BL at Cycle 6 Day 1 | -2.15 (22.69) | -4.39 (20.61) | 0.00 (24.46)
  Change from BL at Cycle 15 or Last Treatment Cycle: number analyzed (Participants) | 142 | 71 | 71
  Change from BL at Cycle 15 or Last Treatment Cycle | -8.45 (25.24) | -8.45 (25.02) | -8.45 (25.65)
  Change from BL at 1.5 Years: number analyzed (Participants) | 146 | 72 | 74
  Change from BL at 1.5 Years | -12.56 (28.27) | -13.89 (30.00) | -11.26 (26.62)
  Change from BL at 2 Years: number analyzed (Participants) | 146 | 73 | 73
  Change from BL at 2 Years | -14.38 (27.93) | -15.98 (27.84) | -12.79 (28.13)
  Change from BL at 3 Years: number analyzed (Participants) | 133 | 68 | 65
  Change from BL at 3 Years | -11.53 (30.99) | -14.71 (32.26) | -8.21 (29.48)

32. Secondary Outcome: Safety Summary for Assessment of Switching Between the FDC SC and IV Formulations: Number of Participants With at Least One Adverse Event During the Treatment Cross-Over Period by Study Arm and Treatment Received
Description: Investigators used the NCI CTCAE v4.0 grading scale for assessing adverse event (AE) severity; if not listed, AE severity was graded as follows: Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe or medically significant; Grade 4 = life-threatening; Grade 5 = death related to AE. Severity and seriousness are not synonymous and investigators independently assessed these criteria for each AE. Investigators also determined whether an AE was considered to be related to the study drug. Adverse events to monitor were defined based on known risks associated with the study drugs and included: hypersensitivity reactions, administration-related reactions (ARRs), cardiac dysfunction, diarrhea grade ≥3, rash/skin reactions, mucositis, interstitial lung disease (ILD), (febrile) neutropenia, pulmonary events that may occur as a result of an ARR, and pregnancy/neonatal related. Multiple occurrences of AEs were counted only once per participant. LVEF = left ventricular ejection fraction
Time Frame: From Day 1 of Cycle 1 to the end of Cycle 3 of Cross-Over Period; from Day 1 of Cycle 4 to the end of Cycle 6 of Cross-Over Period (1 cycle is 21 days)
Population: Safety Population: All participants who received at least one dose of any study treatment categorized according to the study treatment administered. In this analysis, participants are grouped by study arm and treatment received during the Cross-Over Period.
Measure: Count of Participants; unit: Participants
Groups:
- Arm A: Treatment With P+H IV (Cycles 1 to 3): This safety analysis population only includes the adverse events that occurred in Arm A participants during treatment Cycles 1 to 3 when all Arm A participants were treated with P+H IV. In the Treatment Cross-Over Period of the study, participants randomized to Arm A first received treatment with pertuzumab IV and trastuzumab IV (P+H IV) for 3 treatment cycles and that was followed by treatment with pertuzumab and trastuzumab FDC SC (PH FDC SC) for 3 treatment cycles (1 cycle = 21 days).
- Arm A: Treatment With PH FDC SC (Cycles 4 to 6): This safety analysis population only includes adverse events that occurred in Arm A participants during treatment Cycles 4 to 6 when all Arm A participants were treated with PH FDC SC. In the Treatment Cross-Over Period of the study, participants randomized to Arm A first received treatment with pertuzumab IV and trastuzumab IV (P+H IV) for 3 treatment cycles and that was followed by treatment with pertuzumab and trastuzumab FDC SC (PH FDC SC) for 3 treatment cycles (1 cycle = 21 days).
- Arm B: Treatment With PH FDC SC (Cycles 1 to 3): This safety analysis population only includes adverse events that occurred in Arm B participants during treatment Cycles 1 to 3 when all Arm B participants were treated with PH FDC SC. In the Treatment Cross-Over Period of the study, participants randomized to Arm B first received treatment with pertuzumab and trastuzumab FDC SC (PH FDC SC) for 3 treatment cycles and that was followed by treatment with pertuzumab IV and trastuzumab IV (P+H IV) for 3 treatment cycles (1 cycle = 21 days).
- Arm B: Treatment With P+H IV (Cycles 4 to 6): This safety analysis population only includes adverse events that occurred in Arm B participants during treatment Cycles 4 to 6 when all Arm B participants were treated with P+H IV. In the Treatment Cross-Over Period of the study, participants randomized to Arm B first received treatment with pertuzumab and trastuzumab FDC SC (PH FDC SC) for 3 treatment cycles and that was followed by treatment with pertuzumab IV and trastuzumab IV (P+H IV) for 3 treatment cycles (1 cycle = 21 days).
Arm/Group | Arm A: Treatment With P+H IV (Cycles 1 to 3) | Arm A: Treatment With PH FDC SC (Cycles 4 to 6) | Arm B: Treatment With PH FDC SC (Cycles 1 to 3) | Arm B: Treatment With P+H IV (Cycles 4 to 6)
Number analyzed (Participants) | 80 | 80 | 80 | 80
Participants
  Any Adverse Event (AE) | 62 | 60 | 62 | 51
  AE with Fatal Outcome | 0 | 0 | 0 | 0
  Related AE with Fatal Outcome | 0 | 0 | 0 | 0
  Grade 3 to 5 AE | 1 | 1 | 3 | 4
  Related Grade 3 to 5 AE | 1 | 0 | 1 | 0
  Cardiac AE (Including LVEF Events) | 1 | 2 | 3 | 2
  Serious AE | 1 | 1 | 1 | 5
  Anaphylaxis and Hypersensitivity AE, All Grades | 0 | 2 | 1 | 0
  Anaphylaxis and Hypersensitivity AE, Grade ≥3 | 0 | 0 | 0 | 0
  Administration Related Reaction (ARR), All Grades | 7 | 14 | 24 | 2
  Administration Related Reaction (ARR), Grade ≥3 | 0 | 0 | 0 | 0
  Cardiac Dysfunction AE, All Grades | 2 | 1 | 3 | 3
  Cardiac Dysfunction AE, Grade ≥3 | 1 | 0 | 0 | 0
  Diarrhea Grade ≥3 | 0 | 0 | 1 | 0
  Rash/Skin Reactions | 0 | 0 | 0 | 0
  Mucositis | 0 | 0 | 0 | 0
  Pulmonary Events (ARR), All Grades | 18 | 8 | 4 | 8
  Pulmonary Events (ARR), Grade ≥3 | 0 | 0 | 1 | 0
  Pregnancy and Neonatal Related AEs, All Grades | 0 | 0 | 1 | 0
  Pregnancy and Neonatal Related AEs, Grade ≥3 | 0 | 0 | 0 | 0
  Interstitial Lung Disease (ILD) | 0 | 0 | 0 | 0
  Neutropenia/Febrile Neutropenia, All Grades | 4 | 1 | 2 | 3
  Neutropenia/Febrile Neutropenia, Grade ≥3 | 0 | 0 | 0 | 0
  Local Infusion Site Reaction | 1 | 0 | 0 | 0
  Systemic Infusion Site Reaction | 5 | 0 | 0 | 1
  Local Injection Site Reaction | 0 | 12 | 24 | 0
  Systemic Injection Site Reaction | 0 | 2 | 1 | 0
  AE Leading to Any Study Treatment Discontinuation | 0 | 1 | 0 | 0
  AE Leading to PH FDC SC Discontinuation | 0 | 1 | 0 | 0
  AE Leading to Pertuzumab IV Discontinuation | 0 | 0 | 0 | 0
  AE Leading to Trastuzumab IV Discontinuation | 0 | 0 | 0 | 0
  AE Leading to Any Study Treatment Interruption or Dose Reduction | 1 | 0 | 2 | 3

33. Secondary Outcome: Safety Summary of the FDC SC and IV Formulations: Number of Participants With at Least One Adverse Event During the Treatment Cross-Over and Treatment Continuation Periods
Description: as for outcome 32
Time Frame: From Day 1 of Cycle 1 to end of Cycle 6 of the Treatment Cross-Over Period; from Day 1 of Cycle 7 up to the completion of 18 cycles of neo/adjuvant anti-HER2 treatment in the Treatment Continuation Period (1 cycle is 21 days)
Population: Safety Population: All participants who received at least one dose of any study treatment categorized according to the study treatment administered. In this analysis, participants are grouped by treatment received during the Cross-Over and Continuation Periods.
Measure: Count of Participants; unit: Participants
Groups:
- P+H IV: Treatment Cross-Over Period: This safety analysis population includes all participants from Arms A and B who received up to 3 cycles (1 cycle = 21 days) of treatment with pertuzumab IV and trastuzumab IV (P+H IV) during the Treatment Cross-Over Period of the study.
- PH FDC SC: Treatment Cross-Over Period: This safety analysis population includes all participants from Arms A and B who received up to 3 cycles (1 cycle = 21 days) of treatment with the pertuzumab and trastuzumab fixed-dose combination administered subcutaneously (PH FDC SC) during the Treatment Cross-Over Period of the study.
- P+H IV: Treatment Continuation Period: This safety analysis population includes all participants from Arms A and B who, following completion of the Treatment Cross-Over Period, chose to receive pertuzumab IV and trastuzumab IV (P+H IV) during the Treatment Continuation Period for the remaining anti-HER2 treatment cycles (18 planned cycles in total, including pre-study neoadjuvant treatment).
- PH FDC SC: Treatment Continuation Period: This safety analysis population includes all participants from Arms A and B who, following completion of the Treatment Cross-Over Period, chose to receive the pertuzumab and trastuzumab fixed-dose combination administered subcutaneously (PH FDC SC) during the Treatment Continuation Period for the remaining anti-HER2 treatment cycles (18 planned cycles in total, including pre-study neoadjuvant treatment).
Arm/Group | P+H IV: Treatment Cross-Over Period | PH FDC SC: Treatment Cross-Over Period | P+H IV: Treatment Continuation Period | PH FDC SC: Treatment Continuation Period
Number analyzed (Participants) | 160 | 160 | 21 | 138
Participants
  Any Adverse Event (AE) | 113 | 122 | 14 | 92
  AE with Fatal Outcome | 0 | 0 | 0 | 0
  Related AE with Fatal Outcome | 0 | 0 | 0 | 0
  Grade 3 to 5 AE | 5 | 4 | 2 | 7
  Related Grade 3 to 5 AE | 1 | 1 | 0 | 0
  Cardiac AE (Including LVEF Events) | 3 | 5 | 1 | 1
  Serious AE | 6 | 2 | 0 | 4
  Anaphylaxis and Hypersensitivity AE, All Grades | 0 | 3 | 0 | 2
  Anaphylaxis and Hypersensitivity AE, Grade ≥3 | 0 | 0 | 0 | 0
  Administration Related Reaction AE, All Grades | 9 | 38 | 1 | 16
  Administration Related Reaction AE, Grade ≥3 | 0 | 0 | 0 | 0
  Cardiac Dysfunction AE, All Grades | 5 | 4 | 1 | 2
  Cardiac Dysfunction AE, Grade ≥3 | 1 | 0 | 0 | 0
  Diarrhea Grade ≥3 | 0 | 1 | 0 | 0
  Rash/Skin Reactions | 0 | 0 | 0 | 0
  Mucositis | 0 | 0 | 0 | 0
  Pulmonary Events (ARR), All Grades | 26 | 12 | 5 | 13
  Pulmonary Events (ARR), Grade ≥3 | 0 | 1 | 0 | 0
  Pregnancy and Neonatal Related AEs, All Grades | 0 | 1 | 0 | 0
  Pregnancy and Neonatal Related AEs, Grade ≥3 | 0 | 0 | 0 | 0
  Interstitial Lung Disease (ILD), All Grades | 0 | 0 | 0 | 1
  Interstitial Lung Disease (ILD), Grade ≥3 | 0 | 0 | 0 | 0
  Neutropenia/Febrile Neutropenia, All Grades | 7 | 3 | 1 | 5
  Neutropenia/Febrile Neutropenia, Grade ≥3 | 0 | 0 | 0 | 1
  Local Infusion Site Reaction | 1 | 0 | 0 | 0
  Systemic Infusion Site Reaction | 6 | 0 | 1 | 0
  Local Injection Site Reaction | 0 | 36 | 0 | 13
  Systemic Injection Site Reaction | 0 | 3 | 0 | 2
  AE Leading to Any Study Treatment Discontinuation | 0 | 1 | 1 | 0
  AE Leading to PH FDC SC Discontinuation | 0 | 1 | 0 | 0
  AE Leading to Pertuzumab IV Discontinuation | 0 | 0 | 1 | 0
  AE Leading to Trastuzumab IV Discontinuation | 0 | 0 | 1 | 0
  AE Leading to Any Study Treatment Interruption or Dose Reduction | 4 | 2 | 1 | 8

34. Secondary Outcome: Number of Participants With at Least One Event of Heart Failure With the FDC SC and IV Formulations During the Treatment Cross-Over and Treatment Continuation Periods
Description: Heart failure is defined as a disorder characterized by the inability of the heart to pump blood at an adequate volume to meet tissue metabolic requirements, or, the ability to do only at an elevation in the filling pressure. Any adverse event of symptomatic left ventricular systolic dysfunction (LVSD; also referred to as heart failure) occurring during the study was to be reported as a serious adverse event.
Time Frame: as for outcome 33
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | P+H IV: Treatment Cross-Over Period | PH FDC SC: Treatment Cross-Over Period | P+H IV: Treatment Continuation Period | PH FDC SC: Treatment Continuation Period
Number analyzed (Participants) | 160 | 160 | 21 | 138
Participants | 0 | 0 | 0 | 0

35. Secondary Outcome: Number of Participants With at Least One Event of Ejection Fraction Decreased With the FDC SC and IV Formulations During the Treatment Cross-Over and Treatment Continuation Periods
Description: Left ventricular ejection fraction (LVEF) is the measurement of how much blood is being pumped out of the left ventricle of the heart (the main pumping chamber) with each contraction. All participants who enrolled in this study must have had a baseline LVEF ≥55%. Verbatim description of adverse events was mapped to Medical Dictionary for Regulatory Activities (MedDRA) version 25.1. The MedDRA preferred term of 'ejection fraction decreased' is defined as an LVEF decrease of at least 10 percentage points from baseline and to below 50%.
Time Frame: Baseline; Day 1 of Cycles 4, 7, and 11 (each cycle is 21 days); End of Treatment Visit (up to 1 year)
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | P+H IV: Treatment Cross-Over Period | PH FDC SC: Treatment Cross-Over Period | P+H IV: Treatment Continuation Period | PH FDC SC: Treatment Continuation Period
Number analyzed (Participants) | 160 | 160 | 21 | 138
Participants | 3 | 4 | 1 | 0

36. Secondary Outcome: Number of Participants With Targeted Vital Signs Outside the Normal Limits Among Those Without an Abnormality at Baseline During the Treatment Cross-Over and Treatment Continuation Periods
Description: The number of participants at any post-baseline timepoint with abnormal readings outside the normal range for vital signs of diastolic and systolic blood pressure, pulse rate, respiratory rate, and body temperature were summarized according the specified direction of the abnormal reading (high or low). The number analyzed (denominator) in the results table represents participants without the specified abnormal vital sign at baseline. Not every vital sign abnormality qualified as an adverse event (AE). A vital sign result must have been reported as an AE if it met any of the following criteria: was accompanied by clinical symptoms; resulted in a change in study treatment (e.g., dosage modification, treatment interruption, or treatment discontinuation); resulted in a medical intervention or a change in concomitant therapy; or, was clinically significant in the investigator's judgment.
Time Frame: Pre-dose at Day 1 of Cycles 1 (baseline), 4, and 7, and end of treatment (up to 18 cycles; 1 cycle is 21 days)
Population: Safety Population: All participants who received at least one dose of any study treatment categorized according to the study treatment administered. In this analysis, participants are grouped by study arm and treatment received during the Cross-Over Period, and only by treatment received during the Continuation Period. The number analyzed (denominator) represents those without an abnormality at baseline.
Measure: Count of Participants; unit: Participants
Groups:
- Arm A: Treatment With P+H IV (Cycles 1 to 3): This safety analysis population only includes the safety data that was collected from Arm A participants during treatment Cycles 1 to 3 when all Arm A participants were treated with P+H IV. In the Treatment Cross-Over Period of the study, participants randomized to Arm A first received treatment with pertuzumab IV and trastuzumab IV (P+H IV) for 3 treatment cycles and that was followed by treatment with pertuzumab and trastuzumab FDC SC (PH FDC SC) for 3 treatment cycles (1 cycle = 21 days).
- Arm A: Treatment With PH FDC SC (Cycles 4 to 6): This safety analysis population only includes the safety data that was collected from Arm A participants during treatment Cycles 4 to 6 when all Arm A participants were treated with PH FDC SC. In the Treatment Cross-Over Period of the study, participants randomized to Arm A first received treatment with pertuzumab IV and trastuzumab IV (P+H IV) for 3 treatment cycles and that was followed by treatment with pertuzumab and trastuzumab FDC SC (PH FDC SC) for 3 treatment cycles (1 cycle = 21 days).
- Arm B: Treatment With PH FDC SC (Cycles 1 to 3): This safety analysis population only includes the safety data that was collected from Arm B participants during treatment Cycles 1 to 3 when all Arm B participants were treated with PH FDC SC. In the Treatment Cross-Over Period of the study, participants randomized to Arm B first received treatment with pertuzumab and trastuzumab FDC SC (PH FDC SC) for 3 treatment cycles and that was followed by treatment with pertuzumab IV and trastuzumab IV (P+H IV) for 3 treatment cycles (1 cycle = 21 days).
- Arm B: Treatment With P+H IV (Cycles 4 to 6): This safety analysis population only includes the safety data that was collected from Arm B participants during treatment Cycles 4 to 6 when all Arm B participants were treated with P+H IV. In the Treatment Cross-Over Period of the study, participants randomized to Arm B first received treatment with pertuzumab and trastuzumab FDC SC (PH FDC SC) for 3 treatment cycles and that was followed by treatment with pertuzumab IV and trastuzumab IV (P+H IV) for 3 treatment cycles (1 cycle = 21 days).
Arm/Group | Arm A: Treatment With P+H IV (Cycles 1 to 3) | Arm A: Treatment With PH FDC SC (Cycles 4 to 6) | Arm B: Treatment With PH FDC SC (Cycles 1 to 3) | Arm B: Treatment With P+H IV (Cycles 4 to 6) | P+H IV: Treatment Continuation Period | PH FDC SC: Treatment Continuation Period
Number analyzed (Participants) | 80 | 80 | 80 | 80 | 21 | 138
Participants
  Diastolic Blood Pressure - Low: number analyzed (Participants) | 80 | 77 | 80 | 80 | 20 | 137
  Diastolic Blood Pressure - Low | 0 | 0 | 0 | 0 | 0 | 0
  Diastolic Blood Pressure - High: number analyzed (Participants) | 80 | 77 | 78 | 78 | 20 | 135
  Diastolic Blood Pressure - High | 2 | 2 | 0 | 0 | 0 | 3
  Systolic Blood Pressure - Low: number analyzed (Participants) | 80 | 77 | 80 | 80 | 20 | 137
  Systolic Blood Pressure - Low | 0 | 0 | 0 | 0 | 0 | 0
  Systolic Blood Pressure - High: number analyzed (Participants) | 77 | 74 | 75 | 75 | 20 | 129
  Systolic Blood Pressure - High | 8 | 7 | 3 | 3 | 1 | 12
  Pulse Rate - Low: number analyzed (Participants) | 80 | 77 | 80 | 80 | 20 | 137
  Pulse Rate - Low | 0 | 0 | 0 | 0 | 0 | 0
  Pulse Rate - High: number analyzed (Participants) | 75 | 72 | 75 | 75 | 19 | 128
  Pulse Rate - High | 1 | 0 | 0 | 1 | 1 | 1
  Respiratory Rate - Low: number analyzed (Participants) | 80 | 77 | 80 | 79 | 20 | 137
  Respiratory Rate - Low | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory Rate - High: number analyzed (Participants) | 80 | 77 | 79 | 78 | 20 | 136
  Respiratory Rate - High | 1 | 0 | 2 | 2 | 0 | 4
  Temperature - Low: number analyzed (Participants) | 54 | 51 | 39 | 39 | 12 | 80
  Temperature - Low | 22 | 17 | 10 | 13 | 4 | 34
  Temperature - High: number analyzed (Participants) | 80 | 77 | 80 | 80 | 21 | 137
  Temperature - High | 0 | 0 | 1 | 0 | 0 | 0

37. Secondary Outcome: Number of Participants With Chemistry and Hematology Laboratory Test Result Shifts From NCI-CTCAE Grade 0-2 at Baseline to Grade 3-4 Post-Baseline During the Treatment Cross-Over and Treatment Continuation Periods
Description: Laboratory data for targeted chemistry and hematology parameters were classified according to the NCI CTCAE v4.0; Grade 0 is normal and Grades 1 to 4 represent worsening levels of the parameter outside of the normal range in the specified direction of the abnormality (high and low are above and below the range, respectively). The results show the shifts in the number of participants with Grade 0-2 at baseline to Grade 3-4 post-baseline; those with missing baseline values were counted as Grade 0-2 at baseline. Not every laboratory abnormality qualified as an adverse event, only if it met any of the following criteria: was accompanied by clinical symptoms; resulted in a change in study treatment (e.g., dosage modification, treatment interruption, or treatment discontinuation); resulted in a medical intervention or a change in concomitant therapy; or, was clinically significant in the investigator's judgment. SGOT/AST = aspartate aminotransferase; SGPT/ALT = alanine aminotransferase
Time Frame: Pre-dose at Day 1 of Cycles 1 (baseline), 4, 7, 11, 15, and end of treatment (up to 18 cycles; 1 cycle is 21 days)
Population: Safety Population: All participants who received at least one dose of any study treatment categorized according to the study treatment administered. In this analysis, participants are grouped by study arm and treatment received during the Cross-Over Period. The number analyzed (denominator) represents those with NCI-CTCAE Grade 0-2 at baseline and at least one post-baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Treatment With P+H IV (Cycles 1 to 3) | Arm A: Treatment With PH FDC SC (Cycles 4 to 6) | Arm B: Treatment With PH FDC SC (Cycles 1 to 3) | Arm B: Treatment With P+H IV (Cycles 4 to 6) | P+H IV: Treatment Continuation Period | PH FDC SC: Treatment Continuation Period
Number analyzed (Participants) | 80 | 80 | 80 | 80 | 21 | 138
Participants
  Alkaline Phosphatase - High: number analyzed (Participants) | 78 | 79 | 78 | 78 | 21 | 136
  Alkaline Phosphatase - High | 0 | 0 | 0 | 0 | 0 | 0
  SGPT/ALT - High: number analyzed (Participants) | 78 | 79 | 78 | 79 | 21 | 136
  SGPT/ALT - High | 0 | 0 | 0 | 0 | 0 | 0
  SGOT/AST - High: number analyzed (Participants) | 77 | 78 | 79 | 79 | 21 | 136
  SGOT/AST - High | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine - High: number analyzed (Participants) | 80 | 78 | 79 | 77 | 21 | 136
  Creatinine - High | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin, Total - High: number analyzed (Participants) | 76 | 79 | 79 | 79 | 21 | 136
  Bilirubin, Total - High | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin - Low: number analyzed (Participants) | 80 | 78 | 79 | 80 | 21 | 136
  Hemoglobin - Low | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin - High: number analyzed (Participants) | 80 | 78 | 79 | 80 | 21 | 136
  Hemoglobin - High | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils, Total, Abs - Low: number analyzed (Participants) | 80 | 78 | 79 | 80 | 21 | 136
  Neutrophils, Total, Abs - Low | 0 | 0 | 0 | 0 | 0 | 2
  Platelet - Low: number analyzed (Participants) | 80 | 78 | 79 | 80 | 21 | 136
  Platelet - Low | 0 | 0 | 0 | 0 | 0 | 0
  Total Leukocyte Count - Low: number analyzed (Participants) | 80 | 78 | 79 | 80 | 21 | 136
  Total Leukocyte Count - Low | 0 | 0 | 0 | 0 | 0 | 1
  Total Leukocyte Count - High: number analyzed (Participants) | 80 | 78 | 79 | 80 | 21 | 136
  Total Leukocyte Count - High | 0 | 0 | 0 | 0 | 0 | 0

38. Secondary Outcome: Number of Participants With an Event for Overall Survival, Overall and by Treatment Sequence
Description: Overall survival (OS) is defined as the time from randomization to death due to any cause. The number of participants who had an OS event (i.e., died) while on study is reported.
Time Frame: Up to 3 years, 10 months
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 160 | 80 | 80
Participants | 2 | 2 | 0

39. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Were Event-Free for Overall Survival, Overall and by Treatment Sequence
Description: Overall survival is defined as the time from randomization to death due to any cause. Participants who were not reported as having died at the time of analysis were censored at the date when they were last known to be alive. Participants who did not have post-baseline information were censored at the date of randomization +1 day. Kaplan-Meier methodology was used to estimate the percentage of participants who were alive (event-free) at 12, 24, and 36 months.
Time Frame: At 12, 24, and 36 months
Population: ITT Population; the number analyzed at each landmark timepoint represents the number of participants who were remaining at risk for an overall survival event.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 160 | 80 | 80
Percentage of participants
  12 Months: number analyzed (Participants) | 157 | 79 | 78
  12 Months | 100.00 [100.00 to 100.00] | 100.00 [100.00 to 100.00] | 100.00 [100.00 to 100.00]
  24 Months: number analyzed (Participants) | 151 | 76 | 75
  24 Months | 99.36 [98.12 to 100.00] | 98.73 [96.27 to 100.00] | 100.00 [100.00 to 100.00]
  36 Months: number analyzed (Participants) | 97 | 44 | 53
  36 Months | 98.71 [96.92 to 100.00] | 97.44 [93.93 to 100.00] | 100.00 [100.00 to 100.00]

40. Secondary Outcome: Number of Participants With an Event for Invasive Disease-Free Survival Including Second Primary Non-Breast Cancer, Overall and by Treatment Sequence
Description: Invasive Disease-Free Survival is defined as the time from randomization to the first occurrence of one of the following events: ipsilateral invasive breast tumour recurrence, ipsilateral local-regional invasive breast cancer recurrence, distant recurrence, contralateral invasive breast cancer, and death from any cause. Second primary non-breast invasive cancer (with the exception of non-melanoma skin cancers and in situ carcinoma of any site) was included as an event.
Time Frame: Up to 3 years, 10 months
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 160 | 80 | 80
Participants | 12 | 7 | 5

41. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Were Event-Free for Invasive Disease-Free Survival Including Second Primary Non-Breast Cancer, Overall and by Treatment Sequence
Description: Invasive Disease-Free Survival is defined as the time from randomization to the first occurrence of one of the following events: ipsilateral invasive breast tumour recurrence, ipsilateral local-regional invasive breast cancer recurrence, distant recurrence, contralateral invasive breast cancer, and death from any cause. Second primary non-breast invasive cancer (with the exception of non-melanoma skin cancers and in situ carcinoma of any site) was included as an event. Participants who had not experienced invasive disease at the time of analysis were censored: i) at the time of the last clinical breast examination if they had post-baseline clinical breast examination; ii) on the date of randomization +1 day if no post-baseline clinical breast examination. Kaplan-Meier methodology was used to estimate the percentage of participants who were event-free at 12, 24, and 36 months.
Time Frame: At 12, 24, and 36 months
Population: ITT Population; the number analyzed at each landmark timepoint represents the number of participants who were remaining at risk for an invasive-disease free survival (including second primary non-breast cancer) event.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 160 | 80 | 80
Percentage of participants
  12 Months: number analyzed (Participants) | 153 | 75 | 78
  12 Months | 97.46 [95.00 to 99.92] | 94.94 [90.10 to 99.77] | 100.00 [100.00 to 100.00]
  24 Months: number analyzed (Participants) | 143 | 71 | 72
  24 Months | 94.87 [91.40 to 98.33] | 92.37 [86.50 to 98.24] | 97.38 [93.80 to 100.00]
  36 Months: number analyzed (Participants) | 82 | 36 | 46
  36 Months | 93.53 [89.65 to 97.41] | 91.05 [84.72 to 97.38] | 96.03 [91.63 to 100.00]

42. Secondary Outcome: Number of Participants With an Event for Invasive Disease-Free Survival, Overall and by Treatment Sequence
Description: Invasive Disease-Free Survival is defined as the time from randomization to the first occurrence of one of the following events: ipsilateral invasive breast tumour recurrence, ipsilateral local-regional invasive breast cancer recurrence, distant recurrence, contralateral invasive breast cancer, and death from any cause. Ipsilateral or contralateral in situ disease and second primary non-breast cancers (including in situ carcinomas and non-melanoma skin cancers) were not counted as recurrence.
Time Frame: Up to 3 years, 10 months
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 160 | 80 | 80
Participants | 11 | 6 | 5

43. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Were Event-Free for Invasive Disease-Free Survival, Overall and by Treatment Sequence
Description: Invasive Disease-Free Survival is defined as the time from randomization to the first occurrence of one of the following events: ipsilateral invasive breast tumour recurrence, ipsilateral local-regional invasive breast cancer recurrence, distant recurrence, contralateral invasive breast cancer, and death from any cause. Ipsilateral or contralateral in situ disease and second primary non-breast cancers (including in situ carcinomas and non-melanoma skin cancers) were not counted as recurrence. Participants who had not experienced invasive disease at the time of analysis were censored: i) at the time of the last clinical breast examination if they had post-baseline clinical breast examination; ii) on the date of randomization +1 day if no post-baseline clinical breast examination. Kaplan-Meier methodology was used to estimate the percentage of participants who were event-free at 12, 24, and 36 months.
Time Frame: At 12, 24, and 36 months
Population: ITT Population; the number analyzed at each landmark timepoint represents the number of participants who were remaining at risk for an invasive-disease free survival event.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 160 | 80 | 80
Percentage of participants
  12 Months: number analyzed (Participants) | 154 | 76 | 78
  12 Months | 98.10 [95.96 to 100.00] | 96.20 [91.99 to 100.00] | 100.00 [100.00 to 100.00]
  24 Months: number analyzed (Participants) | 144 | 72 | 72
  24 Months | 95.51 [92.25 to 98.76] | 93.64 [88.24 to 99.03] | 97.38 [93.80 to 100.00]
  36 Months: number analyzed (Participants) | 82 | 36 | 46
  36 Months | 94.17 [90.47 to 97.87] | 92.32 [86.41 to 98.23] | 96.03 [91.63 to 100.00]

44. Secondary Outcome: Number of Participants With an Event for Distant Disease-Free Survival, Overall and by Treatment Sequence
Description: Distant disease-free survival (DDFS) is defined as the time from randomization to the date of distant breast cancer recurrence (i.e., evidence of breast cancer in any anatomic site other than for ipsilateral [loco-regional] invasive breast cancer recurrence that has either been histologically confirmed or clinically diagnosed as recurrent invasive breast cancer).
Time Frame: Up to 3 years, 10 months
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 160 | 80 | 80
Participants | 9 | 5 | 4

45. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Were Event-Free for Distant Disease-Free Survival, Overall and by Treatment Sequence
Description: Distant disease-free survival (DDFS) is defined as the time from randomization to the date of distant breast cancer recurrence (i.e., evidence of breast cancer in any anatomic site other than for ipsilateral [loco-regional] invasive breast cancer recurrence that has either been histologically confirmed or clinically diagnosed as recurrent invasive breast cancer). Participants who had not experienced invasive disease at the time of analysis were censored: i) at the time of the last clinical breast examination if they had post-baseline clinical breast examination; ii) on the date of randomization +1 day if no post-baseline clinical breast examination. Kaplan-Meier methodology was used to estimate the percentage of participants who were event-free at 12, 24, and 36 months.
Time Frame: At 12, 24, and 36 months
Population: ITT Population; the number analyzed at each landmark timepoint represents the number of participants who were remaining at risk for a distant disease-free survival event.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants | A: P+H IV Followed by PH FDC SC | B: PH FDC SC Followed by P+H IV
Number analyzed (Participants) | 160 | 80 | 80
Percentage of participants
  12 Months: number analyzed (Participants) | 155 | 77 | 78
  12 Months | 98.73 [96.98 to 100.00] | 97.47 [94.00 to 100.00] | 100.00 [100.00 to 100.00]
  24 Months: number analyzed (Participants) | 145 | 73 | 72
  24 Months | 96.14 [93.11 to 99.17] | 94.90 [90.04 to 99.77] | 97.38 [93.80 to 100.00]
  36 Months: number analyzed (Participants) | 83 | 37 | 46
  36 Months | 94.80 [91.30 to 98.31] | 93.58 [88.14 to 99.03] | 96.03 [91.63 to 100.00]

ADVERSE EVENTS:
Time Frame: AEs and deaths reporting timeframes during study treatment: Cross-Over Period: 3 cycles (cyc) of P+H IV & 3 cyc of PH FDC SC; Continuation Period: from Cyc 7 to 18 total cyc of P+H IV or PH FDC SC (1 cyc = 21 days); All Participants: from first dose through 28 days after last dose of study treatment (up to 1 year). Follow-up period: AEs reported from 29 days up to 7 months after the last dose of study treatment; deaths reported from 29 days after last dose until the end of follow-up (≥3 years).
Description: After initiation of study treatment, all adverse events (AEs) regardless of relationship to study drug were to be reported until 28 days after the last dose of study drug. In the Follow-Up Period, the following AEs were to be reported: study drug-related serious AEs; AEs of special interest, heart failure, pregnancies, non-breast-related second primary malignancies and deaths, irrespective of causal relationship.
Groups:
- PH FDC SC: Treatment Cross-Over Period: This safety analysis population includes all participants from Arms A and B who received up to 3 cycles (1 cycle = 21 days) of treatment with the pertuzumab and trastuzumab fixed-dose combination for subcutaneous administration (PH FDC SC) during the Treatment Cross-Over Period of the study.
- PH FDC SC: Treatment Continuation Period: This safety analysis population includes all participants from Arms A and B who, following completion of the Treatment Cross-Over Period, chose to receive the pertuzumab and trastuzumab fixed-dose combination for subcutaneous administration (PH FDC SC) during the Treatment Continuation Period for the remaining anti-HER2 treatment cycles (18 planned cycles in total, including pre-study neoadjuvant treatment).
- All Participants: All Study Treatment Periods: This safety analysis population includes all participants from Arms A and B who received at least one dose of treatment with pertuzumab IV and trastuzumab IV (P+H IV) and/or the pertuzumab and trastuzumab fixed-dose combination for subcutaneous administration (PH FDC SC) across any of the treatment periods during the study from first dose through 28 days after the last dose of study treatment.
- Follow-Up Period: This safety analysis population includes all participants from Arms A and B who had received at least one dose of any study treatment and had not discontinued from the study prior to entering the follow-up period. The timeframe of the follow-up period started at 29 days after the last dose of study treatment until the end of follow-up (≥3 years after randomization of the last participant).
Arm/Group | P+H IV: Treatment Cross-Over Period | PH FDC SC: Treatment Cross-Over Period | P+H IV: Treatment Continuation Period | PH FDC SC: Treatment Continuation Period | All Participants: All Study Treatment Periods | Follow-Up Period
All-Cause Mortality (participants affected / at risk) | 0/160 | 0/160 | 0/21 | 0/138 | 0/160 | 2/159
Serious Adverse Events (participants affected / at risk) | 6/160 | 2/160 | 0/21 | 4/138 | 11/160 | 1/159
Other Adverse Events (participants affected / at risk) | 62/160 | 84/160 | 10/21 | 47/138 | 125/160 | 2/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | P+H IV: Treatment Cross-Over Period (N=160) | PH FDC SC: Treatment Cross-Over Period (N=160) | P+H IV: Treatment Continuation Period (N=21) | PH FDC SC: Treatment Continuation Period (N=138) | All Participants: All Study Treatment Periods (N=160) | Follow-Up Period (N=159)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0)
Breast cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | P+H IV: Treatment Cross-Over Period (N=160) | PH FDC SC: Treatment Cross-Over Period (N=160) | P+H IV: Treatment Continuation Period (N=21) | PH FDC SC: Treatment Continuation Period (N=138) | All Participants: All Study Treatment Periods (N=160) | Follow-Up Period (N=159)
Diarrhoea (Gastrointestinal disorders) | 17 (20) | 15 (19) | 4 (4) | 15 (23) | 37 (66) | 0 (0)
Fatigue (General disorders) | 8 (8) | 9 (10) | 1 (3) | 7 (8) | 19 (29) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 36 (50) | 0 (0) | 13 (28) | 44 (78) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 27 (29) | 17 (17) | 0 (0) | 1 (1) | 44 (47) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (8) | 8 (9) | 3 (3) | 6 (6) | 23 (26) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3) | 2 (2) | 1 (1) | 12 (12) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 5 (6) | 2 (3) | 1 (1) | 10 (13) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (3) | 3 (3) | 2 (3) | 10 (12) | 0 (0)
Hot flush (Vascular disorders) | 6 (6) | 9 (10) | 0 (0) | 3 (3) | 16 (19) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5) | 2 (2) | 4 (5) | 9 (13) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (8) | 3 (3) | 0 (0) | 7 (7) | 14 (18) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but only after the first publication or presentation that involves the overall study. The Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-12-14): https://cdn.clinicaltrials.gov/large-docs/12/NCT03674112/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/12/NCT03674112/SAP_001.pdf